205883

# TITLE PAGE

**Protocol Title:** A multi-centre, one-arm prospective study to evaluate efficacy and safety of switching from Entecavir (ETV) to Tenofovir Disoproxil Fumarate (TDF) in Japanese chronic hepatitis B HBeAg-positive and HBV-DNA undetectable subjects

**Protocol Number: 205883** 

Short Title: A study of switching from Entecavir to Tenofovir in subjects with chronic hepatitis B

**Compound Number:** GSK548470

# **Sponsor**

GlaxoSmithKline K.K. (GSK)

Akasaka Intercity AIR, 1-8-1, Akasaka, Minato-ku, Tokyo, 107-0052

Person responsible for study implementation:

PPD , VP & Head, Development & Medical Affairs Division

Medical Monitor Name and Contact Information will be provided separately.

Approval Date: [5-Jul-2018]

Copyright 2018 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

| 2017N312381_06 CONFIDENTIAL | 2017N312381_06 | CONFIDENTIAL |
|-----------------------------|----------------|--------------|
|-----------------------------|----------------|--------------|

205883

# **SPONSOR SIGNATORY:**

| [Susie Barnes] | Date |
|-----------------------------------------------------|------|
| [VP & Head, Development & Medical Affairs Division] | |

# TABLE OF CONTENTS

| | | Pa | ıge |
|----|--------------|----------------------------------------------|-----|
| 1. | SYN | OPSIS | 6 |
| 2. | SCH | EDULE OF ACTIVITIES (SOA) | 8 |
| 3. | INT | RODUCTION1 | 2 |
| ; | 3.1. | Study Rationale1 | 2 |
| ; | 3.2. | Background1 | 2 |
| ; | 3.3. | Benefit/Risk Assessment | 2 |
| | 3.3.1 | Risk Assessment1 | 3 |
| | 3.3.2 | 2. Benefit Assessment | 8 |
| | 3.3.3 | 3. Overall Benefit: Risk Conclusion1 | 8 |
| 4. | OBJ | ECTIVES AND ENDPOINTS1 | 8 |
| 5. | STU | DY DESIGN1 | 9 |
| ţ | 5.1. | Overall Design1 | 9 |
| | 5.2. | Number of Subjects1 | 9 |
| ţ | 5.3. | Participant and Study Completion1 | 9 |
| ţ | 5.4. | Scientific Rationale for Study Design | 9 |
| ţ | 5.5. | Dose Justification1 | 9 |
| 6. | STU | DY POPULATION2 | 0 |
| ( | <b>3.1.</b> | Inclusion Criteria | 0 |
| ( | <b>6.2</b> . | Exclusion Criteria2 | 1 |
| ( | 6.3. | Lifestyle Restrictions2 | 2 |
| ( | 6.4. | Screen Failures | 2 |
| 7. | TRE | ATMENT2 | 3 |
| - | 7.1. | Treatments Administered | 3 |
| - | 7.2. | Dose Modification | 3 |
| - | 7.3. | Method of Treatment Assignment | 3 |
| - | 7.4. | Blinding2 | 3 |
| - | 7.5. | Preparation/Handling/Storage/Accountability2 | 4 |
| - | 7.6. | Treatment Compliance | 4 |
| - | 7.7. | Concomitant Therapy2 | 4 |
| - | 7.8. | Treatment after the End of the Study2 | 5 |
| 8. | DISC | CONTINUATION CRITERIA2 | 5 |
| 8 | 3.1. | Discontinuation of Study Treatment | 5 |
| | 8.1.1 | Liver Chemistry Stopping Criteria2 | 5 |
| | 8.1.2 | 2. QTc Stopping Criteria2 | 6 |

| GlaxoSmithKline group of companies |
|------------------------------------|
|------------------------------------|

| | 8.1.3. | | Discontinuation Criteria Related to Renal Function Test Values | 26 |
|---|---|---|---|---|
| | 8.1.4. | | Temporary Discontinuation | 26 |
| 8.1.5. | | 5. | Rechallenge | 26 |
| 8.1.5.1. | | 1.5.1. | Study Treatment Restart or Rechallenge | 26 |
| | 8.1.6 | 6. | Treatment after Discontinuation of Study Treatment | 27 |
| | 8.2. | With | drawal from the Study | |
| | 8.3. | Lost | to Follow Up | 27 |
| 9. | STU | DY A | SSESSMENTS AND PROCEDURES | 28 |
| | 9.1. | Effic | acy Assessments | 28 |
| | 9.1.1 | ١. | Virus test | 28 |
| | 9.1.2 | 2. | Endpoints | 29 |
| | 9.2. | Adve | erse Events | 29 |
| | 9.2.1 | ١. | Time Period and Frequency for Collecting AE and SAE Information | 29 |
| | 9.2.2 | 2. | Method of Detecting AEs and SAEs | |
| | 9.2.3 | 3. | Follow-up of AEs and SAEs | |
| | 9.2.4 | 1. | Regulatory Reporting Requirements for SAEs | |
| | 9.2.5 | 5. | Cardiovascular and Death Events | |
| | 9.2.6 | <b>3</b> . | Disease-Related Events and/or Disease-Related Outcomes Not | |
| | | | Qualifying as SAEs | 31 |
| | 9.2.7 | 7. | Pregnancy | 31 |
| | 9.2.8 | 3. | Medical Device Incidents (Including Malfunctions) | 31 |
| | 9.3. | Trea | tment of Overdose | 31 |
| | 9.4. | Safet | ty Assessments | 31 |
| | 9.4.1 | ١. | Physical Examinations | 32 |
| | 9.4.2 | 2. | Vital Signs | 32 |
| | 9.4.3 | 3. | Electrocardiograms | 32 |
| | 9.4.4 | 1. | Clinical Safety Laboratory Assessments | 32 |
| | 9.4. | 5. | Abdominal Imaging Test | 34 |
| | 9.4.6 | 6. | Bone Densitometry | 34 |
| | 9.5. | Phar | macokinetics | 34 |
| | 9.6. | Phar | macodynamics | 34 |
| | 9.7. | Gene | etics | 34 |
| | 9.8. | Bion | narkers | 34 |
| | 9.9. | Heal | th Economics OR Medical Resource Utilization and Health Economics | 34 |
| 10 | ). STA | TIST | ICAL CONSIDERATIONS | 34 |
| | 10.1. | Samp | ple Size Determination | 34 |
| | 10.1 | .1. | Sample Size Assumptions | 34 |

| 2017N31238 | 81_06 CONFIDENTIAL nKline group of companies 2058 | 02 |
|---|---|---|
| Giaxosiiiili | initine group of companies 2000 | 03 |
| 10.1.2. | . Sample Size Sensitivity3 | 5 |
| 10.1.3. | . Sample Size Re-estimation or Adjustment3 | 5 |
| 10.2. Po | opulations for Analyses3 | 5 |
| 10.3. St | tatistical Analyses3 | 5 |
| 10.3.1. | Efficacy Analyses3 | 6 |
| 10.3.2. | Safety Analyses3 | 6 |
| 10.3.3. | . Interim Analyses3 | 7 |
| 10.3.4. | . Handling of Withdrawed Subjects3 | 7 |
| 11. REFER | RENCES3 | 7 |
| 12. APPEN | NDICES3 | 7 |
| 12.1. A | Appendix 1: Abbreviations and Trademarks3 | 7 |
| 12.2. A | appendix 2: Study Governance Considerations3 | 9 |
| 12.3. A | appendix 3: Adverse Events: Definitions and Procedures for Recording, | |
| E | valuating, Follow-up, and Reporting4 | 3 |
| | appendix 4: Contraceptive Guidance and Collection of Pregnancy | |
| In | nformation4 | 8 |
| | appendix 5: Liver Safety: Required Actions and Follow-up Assessment and | |
| St | tudy Treatment Rechallenge Guidelines5 | 0 |
| 12.6. A | ppendix 6: Prohibited Drugs5 | 3 |
| 12.7. A | ppendix 7: Evaluation of Baseline Values5 | 4 |
| 12.7.1. | Participant Backgrounds5 | 4 |
| 12.7.2. | Diagnosis of Cirrhosis B5 | 4 |
| 12.7.3. | Bone densitometry5 | 4 |

## 1. SYNOPSIS

**Protocol Title:** A multi-centre, one-arm prospective study to evaluate efficacy and safety of switching from Entecavir (ETV) to Tenofovir Disoproxil Fumarate (TDF) in Japanese chronic hepatitis B HBeAg-positive and HBV-DNA undetectable subjects

Short Title: A study of switching from Entecavir to Tenofovir in subjects with chronic hepatitis B

# **Study Rationale:**

This study has been planned to evaluate the virological effects and safety of switching at Day 1 from entecavir hydrate (ETV) to tenofovir disoproxil fumarate (TDF) in chronic hepatitis B HBeAgpositive and HBV-DNA undetectable subjects [ $< 1.3 \log IU/mL$  (< 20 IU/mL) or  $< 2.1 Log_{10}$  copies/mL].

## **Objectives and Endpoints:**

| Objectives | | Endpoints |
|---|---|---|
| Primary | | |
| To evaluate the HBsAg reduction potential a Week 48 | ] | Proportion of subjects achieving 0.25 Log <sub>10</sub> HBsAg reduction from the baseline at Week 48 |
| Secondary | | |
| To evaluate the virological effects | ] | Proportion of subjects achieving 0.25 Log <sub>10</sub> HBsAg reduction from the baseline at Week 24 and 96 |
| | | Proportion of subjects achieving HBsAg loss and HBsAg/Ab seroconversion at Week 24, 48 and 96 |
| | í | Proportion of subjects achieving HBeAg loss and HBeAg/Ab seroconversion at Week 24, 48 and 96 |
| | | Reduction of HBsAg titer from the baseline at Week 24, 48 and 96 |
| | ( | Reduction of HB core-related antigen (HBcrAg) titer from the baseline at Week 24, 48 and 96 |
| To evaluate the safety | • , | Adverse events (AEs) |
| | | Clinical Laboratory values (hematology, clinical chemistry, urinalysis) |
| | 1 | Vital signs (blood pressure, pulse rate, temperature) |
| | • | 12-lead ECG |

| Bone density |
|--------------|
| Done density |

# **Study Design:**

This is a multi-center, one-arm, open-label study. The study will evaluate the efficacy and safety of TDF by switching at Day 1 from ETV to TDF in chronic hepatitis B HBeAg-positive and HBV-DNA undetectable subjects [ $< 1.3 \log IU/mL (< 20 IU/mL)$ or  $< 2.1 Log_{10}$ copies/mL].

# **Number of Subjects:**

Screening, 80 subjects; Subjects eligible for evaluation, 65 subjects

# **Treatment Groups and Duration:**



# 2. SCHEDULE OF ACTIVITIES (SOA)

| Procedure | Screening Treatment period | | | | <b>Discontinuation/Completion</b> | | |
|---|---|---|---|---|---|---|---|
| | (up to 42 | Day 1 | Week 4 | Week 12, | Week 48 | Week 60, 72, 84 | (Week 96) |
| | days | | (±14) | 24, 36 | (±14) | (±14) | $(\pm 14)^2$ |
| | before | | | (±14) | | | |
| | Day 1)1 | | | | | | |
| Informed Consent | $X^1$ | | | | | | |
| Demography | X | | | | | | |
| Abdominal imaging test <sup>3</sup> | X | (X) | (X) | (X) | (X) | (X) | X |
| Inclusion/Exclusion Criteria <sup>4</sup> | X | | | | | | |
| Pregnancy Test (females of childbearing | X | X | X | X | X | X | X |
| potential only ) <sup>5</sup> | | | | | | | |
| [HIV and HCV screening] | X | | | | | | |
| 12-lead ECG | X | | | | X | | X |
| Bone densinometry | $X^6$ | | $(X)^{7,8}$ | $(X)^{7,8}$ | $(X)^{7,8}$ | $(X)^{7,8}$ | $X^8$ |
| Vital Signs <sup>9</sup> | X | X | X | X | X | X | X |
| Study treatment dispensation | | X | | X | X | X | |
| Confirmation of investigational product | | | X | X | X | X | X |
| compliance | | | | | | | |
| AE Assessment | | X | | | | <del> </del> | X |
| SAE Assessment | | X | - | | | <del> </del> | X |
| Concomitant Treatment Review | X | X | 4 | | | <del> </del> - | X |
| Hematology 10 | X | X | X | X | X | X | X |
| Clinical Chemistry 11 | X | X | X | X | X | X | X |
| Urinalysis <sup>12</sup> | X | X | X | X | X | X | X |
| HBV-DNA | X | X | X | X | X | X | X |
| HBeAg/Anti-HBe | X | X | X | X | X | X | X |

| Procedure | Screening | g Treatment period Discontinuation/ | | | | Discontinuation/Completion | |
|---|---|---|---|---|---|---|---|
| | (up to 42<br>days<br>before<br>Day 1) <sup>1</sup> | Day 1 | Week 4<br>(±14) | Week 12,<br>24, 36<br>(±14) | Week 48<br>(±14) | , , | (Week 96)<br>(±14) <sup>2</sup> |
| HBsAg/Anti-HBs | X | X | X | X | X | X | X |
| HBcrAg | | X | X | X | X | X | X |
| Resistant Assay 13 | | | (X) | (X) | (X) | (X) | (X) |
| HBV Genotype | X | | | | | | |

205883

- 1. Perform the screening examinations surely within 42 days before starting the study treatment.
- 2. On completing or discontinuing the study, perform these items within 72 hours after the last dose of the study treatment.
- 3. For diagnosis of cirrhosis, see Appendix 7.
- 4. For subject in whom HBsAg value range is confirmed before screening, enter values at 2 time points (with an interval of at least 3 months, and at least one point within 1 year from screening) into electronic Case Report Form (eCRF).
- 5. Perform the pregnancy test (urine test) for only women of childbearing potential or women with less than two years after the last menstruation. On the day of starting the study treatment, perform the pregnancy test before the first dose of the study treatment.
- 6. If the assessment was performed within 1 year prior to screening, it can be substituted as a score at screening.
- 7. Perform the assessment when the investigator considered necessary from laboratory results.
- 8. Perform bone densimetry with an interval of at least 4 months. If the assessment was performed within 3 months prior to each visit, do not duplicate the procedure.
- 9. Assess height, weight, blood pressure, pulse rate and temperature. Height is collected at screening only.
- 10. Red blood cell count, hemoglobin, hematocrit, white blood cell count (including differential count), platelet count, prothrombin time
- 11. AST, ALT, γ-GTP, ALP, LDH, total bilirubin, direct bilirubin, total protein, serum albumin, serum creatinine, creatinine kinase, amylase, lipase, AFP, antinuclear antibody titer, electrolyte (Na, K, Cl, Ca, P), blood glucose, uric acid, BUN, hyaluronate, lactic acid (however, assess antinuclear antibody titer at screening only, hyaluronate must be assessed at screening but for the visits afterwards assess when necessary), CLcr (calculate from serum creatinine based on Cockcroft-Gault formula described in section 6.1) and eGFR.
- 12. Urinary sediment, β2-microglobulin, urine creatinine, urine glucose, urine protein, electrolyte (P)

# 2017N312381\_06 CONFIDENTIAL

# GlaxoSmithKline group of companies

13. Perform resistance analysis on lamivudine (LAM), adefovir (ADV), ETV and TDF. In a case where a virological breakthrough has been observed (a case where the serum HBV-DNA level has increased from the nadir by at least 1 log IU/mL or an increase of at least 2 log IU/mL (100 IU/mL) if the nadir is under 10 IU/mL), perform the resistance analysis. The blood specimen for the resistance analysis must be taken at every visit (excluding the starting date of the study treatment).

205883

#### 3. INTRODUCTION

Tenofovir Disoproxil Fumarate (TDF) is a nucleos(t)ide analogue that inhibits HBV growth, and is marketed in Japan with an indication for inhibition of HBV growth in patients with chronic hepatitis B associated with HBV growth and abnormal liver function.

CONFIDENTIAL

# 3.1. Study Rationale

This study has been planned to evaluate the virological effects and safety of switching at Day 1 from ETV to TDF in chronic hepatitis B HBeAg-positive and HBV-DNA undetectable subjects.

# 3.2. Background

Chronic hepatitis B (CHB) generally shows exacerbation over a long term by repeating liver inflammation persistently or intermittently. It is known that when chronic hepatitis B is left untreated, liver fibrosis proceeds toward the risk for onset of liver failure or liver cancer [Mizokami, 2010].

There are two options in CHB treatment. One is interferon preparation used by injection and the other is nucleos(t)ide analogue used by oral administration. The interferon therapy does not show a high response rate, since the therapeutic effect is markedly different depending on the initial HBV-DNA level, ALT level and HBV genotype. On the other hand, nucleic acid analogues show a very potent effect to suppress HBV growth, but appearance of HBV strains resistant to each nucleos(t)ide analogue is problematic. Furthermore, the long-term goal of treatment, the loss of HBsAg, is rarely achievable.

It has been reported that TDF demonstrated a superior HBsAg reduction compared to ETV in the Japanese phase 3 study [Koike,2018]. Recently, a topic on the effect of TDF on HBsAg reduction is often seen at conferences in Japan and HBsAg reduction by nucleos(t)ide analogue is drawing attention from the hepatologists. Loss of HBsAg is one of the goals in the 10-year strategy for hepatitis research by the Ministry of Health, Labour and Welfare, and HBsAg is considered an important surrogate marker in CHB treatment.

Based on the above, evaluation of HBsAg reduction in this study is considered medically and clinically significant.

#### 3.3. Benefit/Risk Assessment

More detailed information about the known and expected benefits and risks and reasonably expected adverse events of TDF may be found in the Package Insert.

# 3.3.1. Risk Assessment

2017N312381\_06

| Potential Risk of Clinical Significance | Summary of Data/Rationale for Risk | Mitigation Strategy |
|---|---|---|
| Total Land of Camera Signature | | |
| Renal toxicity | In nonclinical studies, high levels of serum creatinine and chloride, urinary glucose or urinary protein, and increase in urine volume, karyomegaly, denaturation or reproduction, and | Set the inclusion criteria for subjects with creatinine clearance ≥70 mL/min. Set the exclusion criteria for subjects with proximal renal tubular disorders. |
| | necrosis of tubular epithelium, interstitial nephritis, etc. were observed in rats, dogs, and monkeys. The kidney is considered as the target organ of TDF. Although not reported in Japanese clinical studies | Set the dose adjustment when creatinine clearance reaches 50 mL/min. Included prohibited concomitant drugs that affects the kidney. |
| | conducted in subjects infected with HBV, serious renal dysfunction such as renal failure, Fanconi syndrome and other proximal renal tubular disorders have been reported in overseas clinical studies. | Monitor renal function by assessing serum creatinine, etc. during this study period and set the discontinuation criteria based on the renal function values. Collect detailed information on the incidence, |
| | Serious renal dysfunction such as acute renal failure and renal tubular necrosis has been spontaneously reported overseas during the post-marketing use of TDF including preparations with the same ingredients indicated for HIV-1 infection. | seriousness, and outcome of renal toxicity during this study period. |
| | intection. | |

| Potential Risk of Clinical Significance | Summary of Data/Rationale for Risk | Mitigation Strategy |
|---|---|---|
| Bone events (fracture, osteomalacia, etc.) | Effect on serum and urinary phosphorus, range in | Exclude subjects with proximal renal tubular |
| | bone metabolism markers, decrease in bone mineral | disorders through exclusion criteria. |
| | density or bone density, etc. were observed in rats | Monitor serum phosphorus, urinary phosphorus, |
| | and monkeys in non-clinical studies. The bone is | and β2-microglobulin levels, etc. and perform bone |
| | considered the target organ of TDF. | densinometry as necessary, during this study |
| | Tubular epithelium disorder caused by TDF is | period. |
| | considered to lead to a loss of phosphonate into the | Collect detailed information on the incidence, |
| | urine. Accelerated bone resorption associated with | seriousness, and outcome of bone events such as |
| | decreased intestinal absorption of phosphonate is | fracture and osteomalacia during this study period. |
| | also considered responsible for | |
| | bone metabolism disorders leading to bone | |
| | fractures. | |
| | Although not reported in Japanese clinical studies, | |
| | skeletal events such as osteopenia and osteoporosis | |
| | have been reported in overseas clinical studies. | |
| | Fractures and osteomalacia, etc. have been | |
| | spontaneously reported during overseas post- | |
| | marketing use of TDF including preparations with | |
| | the same ingredients indicated for HIV-1 infection. | |

| Potential Risk of Clinical Significance | Summary of Data/Rationale for Risk | Mitigation Strategy |
|---|---|---|
| Hepatic dysfunction (exacerbation of hepatitis after | Hepatitis may occur by regrowth of virus after | Monitor hepatic function by measuring ALT, etc. |
| discontinuation of administration etc) | discontinuation of TDF administration. | during this study period and set the liver chemistry |
| | In the overseas clinical study conducted in subjects | stopping criteria. |
| | infected with HBV, exacerbation of hepatitis at 2-3 | Allow the subjects who meet the stopping criteria |
| | month post treatment discontinuation was observed | and who have been withdrawn from TDF treatment |
| | in 8.75% (7/80 subjects) of the subjects who | can start alternative treatment. |
| | discontinued TDF during the treatment period of up | Collect detailed information on the incidence, |
| | to 240 weeks. | seriousness, and outcome of hepatic dysfunction |
| | Hepatitis flare may occur during oral antiviral | during this study period. |
| | therapy in relation to a rapid decrease of virus, | |
| | characterized by abnormal changes in laboratory | |
| | results such as a rapid elevation of ALT and other | |
| | hepatic function. | |
| Pancreatitis | Increased lipase levels were observed in the | Collect detailed information on the incidence, |
| | Japanese clinical study in subjects infected with | seriousness, and outcome of pancreatitis during this |
| | HBV (2.10%, 3/143 subjects). Also, pancreatitis | study period. |
| | and acute pancreatitis were observed in overseas | |
| | clinical studies. | |
| | Although the incidence is lower than in subjects | |
| | infected with HIV, pancreatitis has been | |
| | spontaneously reported in subjects infected with | |
| | HBV in overseas post-marketing studies. | |

| Potential Risk of Clinical Significance | Summary of Data/Rationale for Risk | Mitigation Strategy |
|---|---|---|
| Lactic acidosis and severe hepatomegaly associated | Lactic acidosis may occur due to the DNA | Collect detailed information on the incidence, |
| with fatty degeneration | polymerase inhibiting function of TDF. | seriousness, and outcome of lactic acidosis and |
| | Occurrence of lactic acidosis has been observed in | severe hepatomegaly associated with |
| | overseas clinical studies of TDF. | fatty degeneration during this study period. |
| | Although the incidence is lower than in subjects | |
| | infected with HIV, lactic acidosis has been | |
| | spontaneously reported in subjects infected with | |
| | HBV in overseas post-marketing studies. | |
| Lipodystrophy | Although not reported in the Japanese or overseas | Collect detailed information on the incidence, |
| | clinical studies in subjects infected with HBV, | seriousness, and outcome of lipodystrophy during |
| | lipodystrophy has been reported in overseas clinical | this study period. |
| | studies in subjects infected with HIV-1. | |
| | Although the incidence is lower than in subjects | |
| | infected with HIV-1, lipodystrophy has been | |
| | spontaneously reported in subjects infected with | |
| | HBV in overseas post-marketing studies. | |
| Drug resistance and cross resistance | Although clinical resistance to TDF has not been | Monitor HBV DNA levels during this study period |
| | confirmed, appearance of TDF-resistant viruses | and perform resistance analysis if virologic |
| | may exacerbate CHB by causing virologic | breakthrough (increase in serum HBV DNA by |
| | breakthrough (rebound of viral load). | ≥1 log IU/mL from the nadir or an increase of at |
| | Although cross-resistance with other drugs has not | least 2 log IU/mL (100 IU/mL) if the nadir is under |
| | been observed in overseas long-term clinical | 10 IU/mL) is observed. |
| | studies of up to 240 weeks, partial cross-resistance | |
| | among HBV reverse transcriptase inhibitors has | |
| | been observed in vitro. | |

| Potential Risk of Clinical Significance | Summary of Data/Rationale for Risk | Mitigation Strategy |
|---|---|---|
| | Study procedures | |
| Change in safety data such as on renal impairment | Although clinical studies conducted overseas | In addition to the mitigation strategy for each of the |
| and change in efficacy data such as on | showed no difference in the change in eGFR levels, | above items, set up a visit at Week 4 to |
| antiviral effect by switching from ETV to TDF | proportion of subjects with a 20% decrease in | obtain/confirm safety and efficacy data at an early |
| | eGFR was reported to be higher in the TDF group | stage after switching to study treatment. |
| | than in the ETV group at Week 96 [Sriprayoon | |
| | 2017]. | |
| | Although clinical resistance to TDF has not been | |
| | confirmed, appearance of TDF-resistant viruses | |
| | may exacerbate CHB by causing virologic | |
| | breakthrough (rebound of viral load). | |

## 3.3.2. Benefit Assessment

In the JSH Guidelines for the Management of Hepatitis B Virus Infection [Drafting Committee for Hepatitis Management Guidelines, the Japan Society of Hepatology 2017], short-term goals of antiretroviral therapy include continuous normalization of ALT level and negative conversion of HBeAg, and short-term goal for subjects on sequential treatment with nucleos(t)ide analogues is negative conversion of HBV DNA. Among these, loss of HBeAg has not been achieved in subjects in this study. As a preliminary step to achieve the long-term goal, HBsAg loss, the decrease in HBsAg level must be observed. However, subjects in this study show high HBsAg levels or no tendency of decrease (fluctuation range of  $\geq$  -0.1 Log<sub>10</sub> IU/mL/year). Since HBsAg reduction was significantly higher in the TDF group compared to the ETV group in the Japanese Phase 3 study [Koike, 2018], switching from ETV to TDF to achieve toward the long-term goal, HBsAg loss, is considered beneficial.

#### 3.3.3. Overall Benefit: Risk Conclusion

Considering the endpoints to minimize risks to the subjects enrolled in the study, the known potential risks of TDF are justified by the potential benefits to CHB subjects.

# 4. OBJECTIVES AND ENDPOINTS

| Objectives | Endpoints |
|---|---|
| Primary | |
| To evaluate the HBsAg reduction potential at Week 48 | <ul> <li>Proportion of subjects achieving 0.25</li> <li>Log<sub>10</sub> HBsAg reduction from the baseline<br/>at Week 48</li> </ul> |
| Secondary | |
| To evaluate the virological effects | <ul> <li>Proportion of subjects achieving 0.25 Log<sub>10</sub> HBsAg reduction from the baseline at Week 24 and 96 </li> <li>Proportion of subjects achieving HBsAg loss and HBsAg/Ab seroconversion at Week 24, 48 and 96</li> <li>Proportion of subjects achieving HBeAg loss and HBeAg/Ab seroconversion at Week 24, 48 and 96</li> <li>Reduction of HBsAg titer from the baseline at Week 24, 48 and 96</li> <li>Reduction of HB core-related antigen (HBcrAg) titerfrom the baseline at Week 24, 48 and 96</li> </ul> |
| To evaluate the safety | Adverse events (AEs) |
| | Clinical laboratory results (hematology,<br>clinical chemistry and urinalysis) |
| | <ul> <li>Vital signs (blood pressure, pulse rate,<br/>temperature)</li> </ul> |
| | • 12-lead ECG |
| | Bone density |

205883

## 5. STUDY DESIGN

# **5.1.** Overall Design



This study is designed as a multi-center, one-arm, post-marketing clinical study. The study will be conducted in CHB HBeAg-positive and HBV-DNA undetectable [< 1.3 log IU/mL (< 20 IU/mL) or < 2.1 Log<sub>10</sub> copies/mL] treated with ETV.

## **5.2.** Number of Subjects

Approximately 80 subjects will be screened to achieve 65 evaluable subjects.

After switching ETV to TDF at Day 1, TDF will be administered for 96 weeks.

## **5.3.** Participant and Study Completion

A subject is considered to have completed the study if he/she has completed all phases of the study including the last visit or the last scheduled procedure shown in the Schedule of Activities (SOA).

The end of the study is defined as the date of the last scheduled procedure shown in the SOA for the last subject in the trial.

## 5.4. Scientific Rationale for Study Design

In this study, on-going ETV treatment is switched to TDF treatment at Day 1 in CHB HBV-DNA undetectable subjects [< 1.3 log IU/mL (< 20 IU/mL) or < 2.1 Log<sub>10</sub> copies/mL]. With regards to the negative conversion of HBV-DNA which is listed as a short-term goal of antiretroviral therapy in the JSH Guidelines for the Management of Hepatitis B Virus Infection, the target subjects are those who are well controlled by ETV treatment. However, as for the negative conversion of HBeAg which is also listed as a short-term goal, the target subjects are those who have not achieved this goal. In addition, this study is designed to investigate the HBsAg reduction in subjects who have not achieved the long-term goal, the loss of HBsAg. The Japanese phase 3 study demonstrated superior HBsAg reduction in TDF treated group compared to the ETV treated group.

The switching of treatment in this study is performed by starting TDF on the day ETV is discontinued, without having overlapping treatment periods. Since both ETV and TDF are oncedaily drugs and the blood concentration of TDF reaches its peak at  $1.2 \pm 0.5$  hr, the method of switching treatment is considered appropriate.

## **5.5.** Dose Justification

As this is a post-marketing clinical study, the dosage and administration of TDF will be 300 mg once daily in accordance with the product package insert.

# **6. STUDY POPULATION**

Prospective approval of protocol deviations to recruitment and enrollment criteria, also known as protocol waivers or exemptions, is not permitted.

# **6.1.** Inclusion Criteria

Subjects are eligible to be included in the study only if all of the following criteria apply:

| Incl | usion Criteria | Screening | Day 1 |
|---|---|---|---|
| 1. | Subjects must be 20 to 69 years of age inclusive, at the time of | X | |
| | signing the informed consent | | |
| 2. | Male and female | X | (X: For |
| | A female subject is eligible to participate if she is not pregnant and | | females, |
| | not breastfeeding (see Appendix 4), and at least one of the | | confirmation |
| | following conditions applies: | | of |
| | | | pregnancy |
| | i) Not a woman of childbearing potential (WOCBP) as | | test only) |
| | defined in Appendix 4 | | |
| | OR | | |
| | ii) A WOCBP who agrees to follow the contraceptive | | |
| | guidance in Appendix 4 during the treatment period and | | |
| | for at least 4 days after the last dose of study treatment | | |
| 3. | Capable of giving signed informed consent form (ICF) as described | X | |
| | in Appendix 2, which includes compliance with the requirements | | |
| | and restrictions listed in the ICF and in this protocol. | | |
| 4. | Subjects with CHB (excluding hospitalized patients) | X | |
| 5. | Subjects treated with ETV for at least 2 years prior to initiation of | | X |
| | study treatment. | | |
| 6. | The serum HBV-DNA level at screening is below the limit of | | X |
| | quantitation [< 1.3 log IU/mL (< 20 IU/mL) or < 2.1 Log <sub>10</sub> | | |
| | copies/mL]. | | |
| 7. | Subjects with serum HBeAg positive at screening | | X |
| 8. | Meet either of the following serum HBsAg levels at screening. | | X |
| | • Serum HBsAg ≥ 800 IU/ml | | |
| | • Serum HBsAg 80 < to < 800 IU/ml | | |
| | and fluctuation decrease is within -0.1 Log <sub>10</sub> IU/ml per year | | |
| | (Confirming the fluctuation range before screening must be | | |
| | determined using the value which has already been measured. | | |
| | Using preserved serum specimen for retest is prohibited.) | | V |
| 9. | Meet all of the following criteria at screening | | X |
| | • Creatinine clearance (CLcr) ≥ 70 mL/min | | |
| | CLcr is calculated using the following Cockcroft-Gault | | |
| | formula. | | |
| | Male: CLcr = (body weight [kg] $\times$ [140-age in years]) / (72 $\times$ | | |
| | serum creatinine [mg/dL]) | | |
| | Female: CLcr = CLcr (male) $\times$ 0.85 | | |
| | • Hemoglobin ≥ 8 g/dL | | |

| • WBC $\geq 1,000 \text{ /mm}^3$ |
|----------------------------------|
|----------------------------------|

# **6.2.** Exclusion Criteria

Subjects are excluded from the study if any of the following criteria apply:

| Exc | lusion Criteria | Screening | Day 1 |
|---|---|---|---|
| 1. | QTc > 450 msec or > 480 msec for subjects with bundle branch | X | |
| | block | | |
| | Note: | | |
| | • QT interval (QTcB) corrected by the Bazett formula, QT | | |
| | interval (QTcF) corrected by the Fridericia formula and/or QT | | |
| | intervals corrected by other formulae. Interpreted by computer | | |
| | or re-interpreted manually. | | |
| | • The QT Interval correction formula used for | | |
| | inclusion/exclusion criteria and discontinuation criteria for | | |
| | each subject should be determined prior to study initiation. | | |
| | Multiple correction formulae cannot be used for QTc | | |
| | calculation for each subject and the lowest QTc value cannot | | |
| | be used for enrolment or discontinuation of subjects. | | |
| 2. | Received any interferon or HB vaccine therapy within 24 weeks | | X |
| | prior to initiation of the study treatment. | | |
| 3. | Received overdose of nonsteroidal anti-inflammatory drugs | | X |
| | (NSAIDs) (excluding temporary or topical use) within 7 days prior | | |
| | to initiation of the study treatment. | | |
| 4. | Received any of the following drugs within 8 weeks prior to | | X |
| | initiation of the study treatment (excluding topical products such as | | |
| | ointment and/or cream etc). | | |
| | • Drugs causing renal impairment (e.g., aminoglycosides, | | |
| | amphotericin B, vancomycin, foscarnet, cisplatin, | | |
| | pentamidine, tacrolimus, cyclosporine, some contrast | | |
| | mediums [ionic high-osmolar contrast media, ionic low- | | |
| | osmolar contrast media] | | |
| | • Competitors of renal excretion (except temporary use, e.g., | | |
| | probenecid) | | |
| | • Immunosuppressants (e.g., azathioprine, cycolphosphamide) | | |
| | or chemotherapeutics (e.g., etoposide) | | |
| | Glucocorticoid preparation | | |
| 5. | Received TDF, ADV or TAF within 2 years prior to initiation of | | X |
| | the study treatment | | |
| 6. | Participation in another clinical study within 6 months prior to | X | |
| | screening, or planned participation in another clinical study | | |
| | simultaneously with this study. | | |
| 7. | Co-infection with HIV or HCV | | X |
| 8. | Subjects with serious complication other than compensated CHB | X | |
| | (cancer, significant renal, cardiovascular, pulmonary, or | | |
| | neurological disease, uncontrollable diabetes, etc.) | | |

| 9. | Received or have a plan for solid organ or bone marrow | X | |
|---|---|---|---|
| ٠. | transplantation | 21 | |
| 10. | Has proximal tubulopathy. | X | |
| 11. | Subjects with decompensated CHB who meet the following. | 11 | X |
| 1 | • Direct bilirubin > 1.5 × ULN, PT < 60%, platelets < | | |
| | 75,000/mm <sup>3</sup> and serum albumin < 3.0 g/dL | | |
| 12. | Diagnosed as an autoimmune hepatitis, excluding CHB | | X |
| 13. | Subjects with or suspected of having hepatocellular carcinoma | | X |
| 13. | (HCC) (including both primary and metastatic) from diagnostic | | A |
| | imaging at screening, or with serum $\alpha$ -fetoprotein (AFP) > 50 | | |
| | ng/mL at screening | | |
| 14. | History of HCC (except subjects who underwent resection or | | X |
| 17. | received curative treatment by radiofrequency, and with AFP $\leq 10$ | | A |
| | ng/mL at screening) | | |
| 15. | Woman who is pregnant, possibly pregnant, lactating or planning a | X | (X: |
| 13. | pregnancy during the study period. | 21 | confirmation |
| | programely during the study portou. | | of |
| | | | pregnancy |
| | | | test only) |
| 16. | Psychiatry disorder or cognitive disorder that may affect the | X | 1020 0223) |
| | subject's ability to give informed consent or to follow specified | | |
| | study procedures. | | |
| 17. | Subjects with a history of alcohol or drug abuse | X | |
| 18. | Subjects whom the investigator (or sub-investigator) considers | X | |
| | ineligible for the study. | | |
| 19. | Subjects with hypersensitivity to study treatments or their | X | |
| | components, nucleoside and/or nucleotide analogues. Subjects with | | |
| | drug allergy that, in the investigator's (sub-investigator's) [or | | |
| | medical monitor's] opinion, labelled contraindication for | | |
| | participation in the study, or other allergy. | | |

## **6.3.** Lifestyle Restrictions

There are no specific lifestyle restrictions in this study.

#### **6.4.** Screen Failures

Screen failures are defined as subjects who consent to participate in the clinical study but are not subsequently entered in the study. A minimal set of screen failure information is required to ensure transparent reporting of screen failure subjects to meet the Consolidated Standards of Reporting Trials (CONSORT) publishing requirements and to respond to queries from regulatory authorities. Minimal information includes demography, screen failure details, eligibility criteria, and any serious adverse events (SAEs).

Information on screen failures as to which participation criteria was not met should be entered into electronic Case Report Form (eCRF) dividing into categories, "failures at screening" and "failures prior to study treatment." For participation criteria to be confirmed at screening and Day 1, refer to Inclusion Criteria and Exclusion Criteria sections.

Individuals who do not meet the criteria for participation in this study (screen failure), regarding to inclusion criteria 4 to 9 or exclusion criteria 2 to 6, may be rescreened for one time only if it is

confirmed that all inclusion criteria are met and exclusion criteria are not met except exclusion criterion 3 after the next visit. There should be an interval of 12 weeks before rescreening. Rescreened subjects should be assigned to the new subject number as from the initial screening.

## 7. TREATMENT

Study treatment is defined as any investigational treatment(s), marketed product(s), placebo, or medical device(s) intended to be administered to a study subject according to the study protocol. The study treatment in this study indicates Tenozet tablet 300 mg as described in Section 7.1.

## 7.1. Treatments Administered

| Study Treatment | Tenofovir Disoproxil Fumarate (Tenozet Tablet 300 mg) |
|---|---|
| Name: | |
| Dosage formulation: | Film-coated tablets |
| Unit dose | 300 mg/dose, once daily |
| strength(s)/Dosage | |
| level(s): | |
| Route of | Oral |
| Administration | |
| Dosing instructions: | 1 tablet per dose |
| Packaging and | A commercially available product, Tenozet Tablets 300 mg, will be used |
| Labeling | for study treatment. |
| Manufacturer: | GlaxoSmithKline K.K. |

#### **7.2.** Dose Modification

In case of CLcr < 50 mL/min, study treatment dose intervals are adjusted in accordance with Table 1:

Table 1 Guidelines for administration corresponding to decreased renal function

| CLcr (mL/min) | Administration method |
|---|---|
| 30 - 49 mL/min | 300 mg once every 2 days |
| 10 - 29 mL/min | 300 mg once every 3-4 days |
| Hemodialysis subjects | 300 mg following dialysis every 7 days <sup>note)</sup> or 300 |
| | mg after a total of approximately 12 hours of |
| | dialysis |

Note) After hemodialysis. Pharmacokinetics in subjects with CLcr <10 mL/minute without hemodialysis has not been evaluated.

## 7.3. Method of Treatment Assignment

There is no randomization in this study.

# 7.4. Blinding

This is an open-label study.

# 7.5. Preparation/Handling/Storage/Accountability

- The study treatment, Tenozet Tablets, will be used from existing stock of the medical institution or dispensed by the medical institution. The sponsor will not provide study treatments.
- 2. Storage and management of study treatment should follow the package insert and procedures of each medical institution.
- 3. Prescription and medication instruction to subjects should follow the procedures of each medical institution.
- 4. The investigator (sub-investigator)/designated staff of the medical institution should document the amount of study treatment dispensed to and the amount taken by subject in the chart (source document).
- Under normal conditions of handling and administration, study treatment is not expected to pose a significant safety risks to the site staff.
- A Material Safety Data Sheet (MSDS)/equivalent document describing occupational hazards
  and recommended handling precautions either will be provided to the investigator, where this
  is required by local laws, or is available upon request from the medical institution.

# **7.6.** Treatment Compliance

• When subjects self-administer study treatment(s) at home, compliance with Tenozet Tablets 300 mg will be assessed through querying the subject during the site visits and documented in the source documents and eCRF. A record of the number of Tenozet Tablets 300 mg dispensed to and taken by each subject must be maintained. Treatment start and stop dates, including those for dose reductions will also be recorded in the eCRF.

## 7.7. Concomitant Therapy

Any medication or vaccine (including over-the-counter or prescription medicines, vitamins, and/or herbal supplements) that the subject is receiving at the time of enrolment or receives during the study must be recorded along with:

- reason for use
- dates of administration including start and end dates
- dosage information including dose and frequency

The Medical Monitor should be contacted if there are any questions regarding concomitant or prior therapy.

### Permitted Concomitant Drugs

Appendix 6: Drug not specified in "Prohibited Drugs" may be used concomitantly. However, on using the following drugs concomitantly, the instructions shown below should be taken into consideration. It is permitted to use a contrast medium considered less influential on the kidney, only in a case where an imaging test by CT or MRI needing a contrast medium is clinically necessary in order not to miss the onset of liver cancer.

Non- ionic low osmolar contrast media, contrast media for MRI

Note: Each contrast medium should be administered carefully paying attention to the renal functions by, e.g., securing the urine amount with transfusion of physiological saline before and

205883

after using the contrast medium as the measures to prevent renal impairment of the contrast medium. Furthermore, more careful administration is necessary in case of using the contrast medium in subjects with decreased renal function.

#### **Prohibited Concomitant Drugs**

During the period from the start to completion of study treatment, concomitant use of the drugs listed in "Appendix 6: Prohibited drugs" will be prohibited due to the possibility of having the impact on efficacy and safety evaluation.

However, the following drug, which is listed in "Appendix 6: Prohibited drugs," may be used for the purpose of liver supporting therapy.

#### 1. Ursodeoxycholic acid preparations

When the ALT or AST level exceeds 10 times the ULN, rescue medication may be used after consultation with the medical monitor of the sponsor. Rescue medication name, date administered, and administration method must be documented.

## 7.8. Treatment after the End of the Study

After the completion of study treatment and subject's last visit, the investigator (sub-investigator) will perform the treatment considered most appropriate for each subject. The investigator (sub-investigator) is responsible for considering the subject's medical care whether or not the sponsor provides specific treatment after study completion.

## 8. DISCONTINUATION CRITERIA

# **8.1.** Discontinuation of Study Treatment

# **8.1.1.** Liver Chemistry Stopping Criteria

**Liver chemistry stopping and increased monitoring criteria** have been designed to assure subject safety and evaluate liver event etiology.

If a subject corresponds to any of the following conditions, discontinuation of study treatment due to abnormal liver function test result is required.

- When a subject corresponds to any of the following conditions
  - Bilirubin  $\geq 2$  times ULN and direct bilirubin  $\geq 35\%$
  - International Normalized Ratio (INR) > 1.5 without the administration of warfarin
  - Evidence of clinical liver decompensation (development of encephalopathy, ascites, hypoalbuminemia [albumin ≤ 3 g/dL]) or variceal bleeding
  - ALT ≥ 20 times ULN in the absence of increased bilirubin or evidence of clinical decompensation, if persisting ≥ 2 weeks or accompanied by worsening hepatitis symptoms.

OR

The investigator (sub-investigator) considered it to be in the best interest of the subject to discontinue study treatment, although the abnormal liver function test values of the subject do not meet the criteria for discontinuation specified in the protocol.

Required actions after liver event and the follow-up assessment section are shown in Appendix 5.

## 8.1.2. QTc Stopping Criteria

- The same QT correction formula must be used for each individual subject to determine eligibility for and discontinuation from the study. This formula may not be changed or substituted once the subject has been enrolled.
  - For example, if a subject is eligible for the protocol based on QTcB, then QTcB must be used for discontinuation of this individual subject as well.
  - Once the QT correction formula has been chosen for a subject's eligibility, the same formula must continue to be used for that subject for all QTc data being collected for data analysis. Safety ECGs and other non-protocol specified ECGs are an exception.
- The QTc should be based on single ECG.

If ECG results show the following, the subject should be withdrawn from the study.

• QTc > 500 msec or uncorrected QT > 600 msec

For subjects with bundle branch block, the following stopping criteria should be followed.

| Baseline value in subjects with bundle branch block | Stopping criteria in subjects with bundle |
|---|---|
| | branch block |
| < 450 msec | > 500 msec |
| 450 - 480 msec | ≥530 msec |

See the SOA for data to be collected at the time of treatment discontinuation of study and followup and for any further evaluations that need to be completed.

#### 8.1.3. Discontinuation Criteria Related to Renal Function Test Values

The discontinuation criteria and follow-up observation criteria related to renal function test values will be specified in order to secure the safety of the subjects.

Serum creatinine values  $\geq 0.5$  mg/dL above baseline should be confirmed by repeat testing within 3 calendar days of receipt of results before the study treatment is discontinued. (However, if such a delay of study treatment discontinuation concerns the safety of subject, study treatment should be discontinued immediately.) For serum creatinine elevation  $\geq 0.5$  mg/dL above baseline, subjects may continue all study medication, but it is recommended that subjects should be monitored weekly until the serum creatinine returned to the original baseline value or  $\leq 0.3$  mg/dL from baseline.

All study treatments should be permanently discontinued in the event that repeated testing of serum creatinine confirms > 2 mg/dL. The subject should be followed weekly until the serum creatinine reaches within 0.3 mg/dL elevation of the baseline value.

## **8.1.4.** Temporary Discontinuation

Subjects who stopped study treatment will be withdrawn from this study.

# 8.1.5. Rechallenge

## **8.1.5.1.** Study Treatment Restart or Rechallenge

Study treatment restart or rechallenge is not allowed if study subject meets any of the stopping criteria specified in each section under 8.1.

# 8.1.6. Treatment after Discontinuation of Study Treatment

Subjects who meet stopping criteria and who have been withdrawn from study treatment can start alternative treatment.

# 8.2. Withdrawal from the Study

If one of the following events 1) to 6) occurs in a subject, the investigator (or sub-investigator) should withdraw that subject from the study:

- 1) When the subject is lost to follow-up.
- 2) When the subject or subject's legally acceptable representative wishes to withdraw from the study.
- 3) When it is confirmed that the subject is pregnant.
- 4) When the subject meets QTc stopping criteria (refer to 8.1.2. QTc stopping criteria).
- 5) When the subject stopping criteria related to hepatic or renal function test values (refer to 8.1.1. Liver Chemistry Stopping Criteria or 8.1.3. Discontinuation Criteria Related to Renal Function Test Values).
- 6) When the study is prematurely terminated for other reasons not directly related to the study

If one of the following events 7) to 11) occurs in asubject, the investigator (or sub-investigator) may, at their discretion, withdraw that subject from the study:

- 7) When it is difficult to continue the study due to an adverse event (s) (Refer to the package insert of Tenozet Tablets 300 mg).
- 8) When a protocol deviation is found
- 9) When it is difficult to continue the study due to exacerbation of the primary disease or a complication
- 10) When the disease being studied resolved
- 11) When the investigator (or sub-investigator) considers necessary to withdraw the subject from the study for other reasons.

If one of the following events 1) to 11) occurs, reason for withdrawal and date of withdrawal should be entered into eCRF while taking necessary measures. If the consent is withdrawed, the reason must be entered into eCRF.

- A subject may withdraw from the study at any time at his/her own request, or may be withdrawn at any time at the discretion of the investigator for safety, behavioral, compliance or administrative reasons.
- If the subject withdraws consent for disclosure of future information, the sponsor may retain and continue to use any data collected before such a withdrawal of consent.
- If a subject withdraws from the study, he/she may request destruction of any samples taken and not tested, and the investigator must document this in the site study records.
- Refer to the SOA for data to be collected at the time of study discontinuation and follow-up and for any further evaluations that need to be completed.

# 8.3. Lost to Follow Up

A subject will be considered lost to follow-up if he or she repeatedly fails to return for scheduled visits and is unable to be contacted by the study site.

The following actions must be taken if a subject fails to return to the clinic for a required study visit:

- The site must attempt to contact the subject and reschedule the missed visit as soon as possible and counsel the subject on the importance of maintaining the assigned visit schedule and ascertain whether or not the participant wishes to and/or should continue in the study.
- Before a subject is deemed lost to follow up, the investigator or designee must make every effort to regain contact with the subject (where possible, 3 telephone calls and, if necessary, a certified letter to the subject's last known mailing address or local equivalent methods). These contact attempts should be documented in the subject's medical record.
- Should the subject continue to be unreachable, he/she will be considered to have withdrawn from the study with a primary reason of lost to follow-up.

# 9. STUDY ASSESSMENTS AND PROCEDURES

- Study procedures and their timing are summarized in the SOA.
- Protocol waivers or exemptions are not allowed.
- Immediate safety concerns should be discussed with the sponsor immediately upon occurrence or awareness to determine if the subject should continue or discontinue study treatment.
- Adherence to the study design requirements, including those specified in the SOA, is essential and required for study conduct.
- All screening evaluations must be completed and reviewed to confirm that potential subjects
  meet all eligibility criteria. The investigator will maintain a screening log to record details of
  all subjects screened and to confirm eligibility or record reasons for screening failure, as
  applicable.
- Procedures conducted as part of the subject's routine clinical management (e.g., blood count)
  and obtained before signing of ICF may be utilized for screening or baseline purposes
  provided the procedure met the protocol-specified criteria and was performed within the time
  frame defined in the SOA.
- Repeat or unscheduled samples may be taken for safety reasons or for technical issues with the samples.

# **9.1.** Efficacy Assessments

## **9.1.1.** Virus test

According to the SOA, the following virus tests will be performed on the specified days. These tests will be performed centrally at SRL Inc. in principle. The test results will be reported to each study site and the sponsor.

- HIV, HCV (only at the time of screening)
- HBV Genotype (only at the time of screening)
- HBV-DNA levels (at screening, Day 1 of administration, Week 4, every 12 weeks)
- HBe Ag/Ab, HBs Ag/Ab (quantitation) (at the time of screening, Day 1 of administration, Week 4, every 12 weeks)
- HB cr Ag (Day 1 of administration, Week 4, every 12 weeks)
- LAM resistance analysis, ADV resistance analysis, ETV resistance analysis, TDF resistance analysis (a case where the serum HBV-DNA level has increased from the nadir by at least 1 log IU/mL or an increase of at least 2 log IU/mL (100 IU/mL) if the nadir is under 10 IU/mL)

The blood sample for the resistance analysis should surely be taken at each visit and the resistance analysis will be performed in the above cases. Blood samples taken for resistance analysis will be stored at SRL Inc. until completion of study.

## 9.1.2. Endpoints

#### **Primary Endpoint**

Proportion of subjects achieving 0.25 Log<sub>10</sub> HBsAg reduction from the baseline at Week 48

## **Secondary Endpoints**

- 1. Proportion of subjects achieving 0.25 Log<sub>10</sub> HBsAg reduction from the baseline at Week 24 and 96
- 2. Proportion of subjects achieving HBsAg loss and HBsAg/Ab seroconversion at Week 24, 48 and 96
- 3. Proportion of subjects achieving HBeAg loss and HBeAg/Ab seroconversion at Week 24, 48 and 96
- 4. Reduction of HBsAg titer from the baseline at Week 24, 48 and 96
- 5. Reduction of HBcrAg titer from the baseline at Week 24, 48 and 96

#### 9.2. Adverse Events

The definitions of an AE or SAE can be found in Appendix 3.

The investigator and any designees are responsible for detecting, documenting, and reporting events that meet the definition of an AE or SAE and remain responsible for following up AEs that are serious, considered related to the study treatment or the study, or that caused the subject to discontinue the study treatment (see Section 8).

# **9.2.1.** Time Period and Frequency for Collecting AE and SAE Information

- All SAEs will be collected from the start of study treatment until completion/discontinuation
  of study at the time points specified in the SOA (Section 2). However, study participation
  (e.g., study treatment, procedures specified in the protocol, invasive testing, or change from
  the current therapy) or all SAEs considered associated with GSK products will be recorded
  from the time the subjectgave consent to participation in the study.
- All AEs will be collected from the start of treatment until completion/discontinuation of the study at the time points specified in the SOA (Section 2).
- Medical occurrences that begin before the start of study treatment but after obtaining informed consent will be recorded on the Medical History/Current Medical Conditions section of the case report form (CRF) not the AE section.
- All SAEs will be recorded and reported immediately, but no longer than 24 hours in any
  circumstances, to the sponsor or designee as indicated in Appendix 3. The investigator (subinvestigator) will submit any updated SAE data to the sponsor within 24 hours of it being
  available.
- Investigators (sub-investigators) are not obligated to actively seek AEs or SAEs in former study subjects. However, if the investigator learns of any SAE, including a death, at any time after a subjecthas been discharged from the study, and he/she considers the event to be reasonably related to the study treatment or study participation, the investigator must promptly notify the sponsor.

- The method of recording, evaluating, and assessing causality of AEs and SAEs and the procedures for completing and transmitting SAE reports are provided in Appendix 3.
- All non-serious AEs considered associated with the study treatment in the post-marketing clinical study will be recorded and reported to the sponsor or designee within 24 hours of it being available as indicated in Appendix 3.

# 9.2.2. Method of Detecting AEs and SAEs

Care will be taken not to introduce bias when detecting AE and/or SAE. Open-ended and non-leading verbal questioning of the subjectis the preferred method to inquire about AE occurrence.

# 9.2.3. Follow-up of AEs and SAEs

After the initial AE/SAE report, the investigator is required to proactively follow each subjectat subsequent visits/contacts. All SAEs will be followed until the event is resolved, stabilized, otherwise explained, or the subjectis lost to follow-up (as defined in Section 8.3). Further information on follow-up procedures is given in Appendix 3.

Non-serious AEs considered associated with the study treatment in the post-marketing clinical study will also be followed.

# 9.2.4. Regulatory Reporting Requirements for SAEs

- Prompt notification by the investigator to the sponsor of an SAE is essential so that legal
  obligations and ethical responsibilities towards the safety of subjects and the safety of a study
  treatment under clinical investigation are met.
- The sponsor has a legal responsibility to notify both the local regulatory authority and other
  regulatory agencies about the safety of a study treatment under clinical investigation. The
  sponsor will comply with country-specific regulatory requirements relating to safety
  reporting to the regulatory authority, Institutional Review Boards (IRB)/Independent Ethics
  Committees (IEC), and investigators.
- Investigator safety reports must be prepared for suspected unexpected serious adverse reactions (SUSAR) according to local regulatory requirements and sponsor policy and forwarded to investigators as necessary.
- An investigator who receives an investigator safety report describing a SAE or other specific safety information (e.g., summary or listing of SAE) from the sponsor will review and then file it along with the Investigator's Brochure and will notify the IRB/IEC, if appropriate according to local requirements.
- Prompt notification to the sponsor of non-serious AEs considered associated with the study
  treatment in post-marketing clinical study is essential so that legal obligations and ethical
  responsibilities towards the safety of subjects and the safety of a study treatment under
  clinical investigation are met.

## **9.2.5.** Cardiovascular and Death Events

For any cardiovascular events detailed in Appendix 3 and all deaths, whether or not they are considered SAEs, specific Cardiovascular (CV) and Death sections of the CRF will be required to be completed. These sections include questions regarding cardiovascular (including sudden cardiac death) and non-cardiovascular death.

#### 205883

The CV CRFs are presented as queries in response to reporting of certain CV MedDRA terms. The CV information should be recorded in the specific cardiovascular section of the CRF within one week of receipt of a CV Event data query prompting its completion.

The Death CRF is provided immediately after the occurrence or outcome of death is reported. Initial and follow-up reports regarding death must be completed within one week of when the death is reported.

# **9.2.6.** Disease-Related Events and/or Disease-Related Outcomes Not Qualifying as SAEs Not applicable

# 9.2.7. Pregnancy

- Details of all pregnancies in female subjects will be collected after the start of study treatment until 4 days after the last dose.
- If a pregnancy is reported, the investigator (sub-investigator) should inform GSK within 24 hours of learning of the pregnancy and should follow the procedures outlined in Appendix 4.
- Abnormal pregnancy outcomes (e.g., spontaneous abortion, fetal death, stillbirth, congenital anomalies, ectopic pregnancy) are considered SAEs.

# **9.2.8.** Medical Device Incidents (Including Malfunctions)

Not applicable

#### **9.3.** Treatment of Overdose

For this study, any dose of TDF greater than 300 mg within a 1-day period will be considered an overdose.

The package insert of TDF (Tenozet Tablets 300 mg) describes overdose as follows.

No case of overdose of TDF has been reported and specific signs and symptoms at the time of overdose are unknown. Closely monitor the subjectfor adverse reactions to TDF at the time of overdose and perform symptomatic therapy as needed. TDF can partially be removed by hemodialysis. Tenofovir removal by peritoneal dialysis has not been examined.

In the event of an overdose, the investigator (sub-investigator) should:

- 1. Contact the Medical Monitor immediately.
- 2. Closely monitor the subject for AE/SAE and laboratory abnormalities until Tenofovir can no longer be detected (at least 4 days).
- 3. Obtain a plasma sample for PK analysis within 24 hours from the date of the last dose of study treatment if requested by the Medical Monitor (determined on a case-by-case basis).
- 4. Document the quantity of the excess dose as well as the duration of the overdosing in the CRF.

Decisions regarding dose interruptions or modifications will be made by the investigator (sub-investigator) in consultation with the sponsor's Medical Monitor based on the clinical evaluation of the subject.

# 9.4. Safety Assessments

Planned time points for all safety assessments are provided in the SOA.

#### **9.4.1.** Physical Examinations

- A complete physical examination will include, at a minimum, assessments of the Skin, Cardiovascular, Respiratory, Gastrointestinal and Neurological systems. Height and weight will also be measured and recorded.
- A brief physical examination will include, at a minimum, assessments of the skin, lungs, cardiovascular system, and abdomen (liver and spleen).
- Investigator (sub-investigator) should pay special attention to clinical signs related to previous serious illnesses.

# 9.4.2. Vital Signs

- Temperature (axillary), pulse rate, and blood pressure will be assessed.
- Blood pressure and pulse measurements will be assessed with a completely automated device. Manual techniques will be used only if an automated device is not available.
- Blood pressure and pulse measurements should be preceded by at least 5 minutes of rest for the subjectin a quiet setting without distractions (e.g., television, cell phones).
- Vital signs (to be taken before blood collection for laboratory tests) will consist of 1 pulse and 3 blood pressure measurements (3 consecutive blood pressure readings will be recorded at intervals of at least 1 minute). The average of the 3 blood pressure readings will be recorded on the CRF.

# 9.4.3. Electrocardiograms

- Single 12-lead ECG will be obtained as outlined in the SOA (Section 2) at screening, Week 48, at discontinuation or completion of study, and that automatically calculates the heart rate and measures PR, QRS, QT, and QTc intervals. Refer to Section 8.1.2 for QTc withdrawal criteria and additional QTc readings that may be necessary.
- The measured ECG Waveforms will be retained at each medical institution in paper or electronic form.

# 9.4.4. Clinical Safety Laboratory Assessments

- Refer to Table 2 for the list of clinical laboratory tests to be performed and to the SOA for the timing and frequency.
- The investigator (sub-investigator) must review the laboratory report, document this review, and record any clinically relevant changes occurring during the study in the AE section of the CRF. The laboratory reports must be filed with the source documents. Clinically significant abnormal laboratory findings are those which are not associated with the underlying disease, unless judged by the investigator (sub-investigator) to be more severe than expected for the subject's condition.
- All laboratory tests with values considered clinically significantly abnormal during
  participation in the study or within 4 days after the last dose of study treatment should be
  repeated until the values return to normal or baseline or are no longer considered
  significantly abnormal by the investigator or medical monitor.
- If such values do not return to normal/baseline within a period of time judged reasonable by the investigator, the etiology should be identified and the sponsor notified.
- All protocol-required laboratory assessments, as defined in Table 2, must be conducted in accordance with the laboratory manual and the SOA.
- The laboratory tests detailed in Table 2 will be performed by the central laboratory.

 Protocol-specific inclusion/exclusion criteria for subjects are included in Section 6 of the protocol.

CONFIDENTIAL

• Additional tests may be performed at any time during the study as determined necessary by the investigator (sub-investigator) or required by local regulations.

**Table 2** Protocol-Required Safety Laboratory Assessments

| Laboratory | Parameters | | | | | |
|---|---|---|---|---|---|---|
| Assessments | - m.m | | | | | |
| Hematology | Platelet Count Hemoglobin | | | | WBC count with | |
| | | | | | Differential: | |
| | | | | | Neutrophils | |
| | | | | | Lymp | phocytes |
| | | | | Mono | | cytes |
| | | | | | Eosino | ophils |
| | | | | | Basophils | |
| | RBC Count | | Hematocrit | | Prothr | ombin time |
| Clinical | Blood urea | LDH | | Aspartate | • | Total and direct |
| Chemistry <sup>1</sup> | nitrogen (BUN) | | | Aminotransfe | erase | bilirubin |
| | | | | (AST)/ Serur | n | |
| | | | | Glutamic- | | |
| | | | | Oxaloacetic | | |
| | | | | Transaminase | | |
| | | | | (SGOT) | | |
| | Creatinine | CLcr | | Alanine | | Total Protein |
| | | | | Aminotransferase | | |
| | | | | (ALT)/ Serum | | |
| | | | | Glutamic-Pyruvic | | |
| | | | | Transaminase | | |
| | | | | (SGPT) | | |
| | Glucose [fasting | eGFR | | Alkaline | | γ-GTP |
| | not required] | | | phosphatase | (ALP) | |
| | Albumin | Creati | ne kinase | Amylase | | Lipase |
| | AFP | Antinu | uclear | Electrolyte (1 | Na, K, | Uric acid |
| | | antibo | dy titer [only | Cl, Ca, P) | | |
| | | at the | time of | | | |
| | | screening] Lactic Acid | | | | |
| | Hyaluronic acid | | | | | |
| | [Required at | | | | | |
| | screening and as | | | | | |
| | needed thereafter.] | | | | | |
| Urinalysis | | | <u> </u> | | | nt, β2-microglobulin |
| Other screening | | | | | | |
| tests | childbearing potential and if required) <sup>2</sup> | | | | | |

# Notes:

1. Details of liver chemistry stopping criteria, required actions after liver events and follow-up assessments are provided in Section 8.1 and Appendix 5.

2. Local urine testing will be standard for the protocol unless serum testing is required by local regulation or IRB/IEC.

# 9.4.5. Abdominal Imaging Test

Abdominal imaging test will be performed to diagnose HCC and hepatic cirrhosis in accordance with the SOA (Section 2).

# **9.4.6.** Bone Densitometry

Bone densitometry will be performed using DEXA, SEXA, or ultrasound in accordance with the SOA (Section 2). Refer to Appendix 7.

#### 9.5. Pharmacokinetics

PK parameters are not evaluated in this study.

## 9.6. Pharmacodynamics

Pharmacodynamic parameters are not evaluated in this study.

#### 9.7. Genetics

Genetics are not evaluated in this study.

#### 9.8. Biomarkers

Biomarkers are not evaluated in this study.

#### 9.9. Health Economics OR Medical Resource Utilization and Health Economics

Health Economics/Medical Resource Utilization and Health Economics parameters are not evaluated in this study.

# 10. STATISTICAL CONSIDERATIONS

This is an open-label uncontrolled study to evaluate the virological effects and safety of switching at Day 1 from ETV to TDF 300 mg once daily in Japanese CHB HBeAg-positive and HBV-DNA undetectable subjects [ $< 1.3 \log IU/mL (< 20 IU/mL)$ or  $< 2.1 Log_{10}$ copies/mL]. Exploratory investigation will therefore be performed and no confirmatory hypotheses will be tested. Descriptive summary will be used to assess the efficacy and safety objectives.

# **10.1.** Sample Size Determination

## **10.1.1.** Sample Size Assumptions

Although no confirmatory hypotheses will be tested in this study, the sample size has been examined using the expected responder rate and threshold rate. Assuming the proportion of subjects achieving 0.25 Log<sub>10</sub> HBsAg reduction from the baseline (proportion of HBsAg responder) at Week 48 to be 20%, the proportion of HBsAg responder in subjects not switched to TDF-based regimens on the basis of results of ETV treatment to be 6% (threshold rate), and significance level (two tailed) to be 5%, the sample size with at least 90% power is calculated to be 57. Allowing for a dropout rate of 10%, the sample size is calculated to be 64 and thus the target sample size was set at approximately 65.

# **10.1.2.** Sample Size Sensitivity

Table 3 shows the sample sizes needed to have an at least 80% or 90% power, assuming a 15% to 25% expected proportion of subjects achieving 0.25 Log<sub>10</sub> HBsAg reduction from the baseline and a 6% to 10% threshold proportion of subjects.

 Table 3
 Sample size calculation

| Threshold (%) | The proportion of | $\geq$ 80% power (N) | $\geq$ 90% power (N) |
|---|---|---|---|
| | HbsAg responder at | | |
| | Week 48 (%) | | |
| 6 | 15 | 82 | 116 |
| | 20 | 55 | 57 |
| | 25 | 55 | 55 |
| 8 | 15 | 156 | 215 |
| | 20 | 61 | 86 |
| | 25 | 40 | 45 |
| 10 | 15 | 341 | 455 |
| | 20 | 94 | 132 |
| | 25 | 49 | 64 |

# 10.1.3. Sample Size Re-estimation or Adjustment

No sample size re-estimation will be performed.

# **10.2.** Populations for Analyses

For analysis purposes, the following populations are defined:

| Population | Description |
|---|---|
| Enrolled | Subjects who provided consent |
| Screen failures | Subjects who provided consent but were not subsequently |
| | administered |
| Safety Population: SP | Subjects who have received at least 1 dose of study treatment after |
| | enrolment. |
| Full Analysis Set: FAS | A population of all subjects enrolled in the study, excluding those |
| | who meet either of the following criteria. |
| | Have not received any dose of study treatment. |
| | Have no efficacy data after the start of study treatment. |
| Efficacy Evaluable Set: | A subset of subjects in the FAS defined above and evaluable for |
| EES | efficacy. |
| | Refer to Report and analysis plan (RAP) for more details. |

# 10.3. Statistical Analyses

The data in this study will be presented in the form of tables and/or graphs and descriptively summarized in accordance with the Integrated Data Standards Library (IDSL) of the sponsor (GSK).

Detailed analyses will be described in the Report and analysis plan (RAP).

#### **10.3.1.** Efficacy Analyses

Efficacy analyses will be performed on the FAS. Primary endpoint analyses will be performed also on EES.

#### Statistical methods

The primary endpoint is the proportion of subjects achieving 0.25 Log<sub>10</sub> HBsAg reduction from the baseline at Week 48, and the responder rate and its two-sided 95% confidence interval will be calculated.

As the secondary analysis, the responder rate (%) at Week 24 and Week 96 and its two-sided 95% confidence interval will also be calculated.

Analyses similar to the primary analysis will also be performed in subgroups (disease, genotype, etc.). These subgroup analyses are intended to assess the robustness of results.

#### Subgroup:

- Disease (CHB, liver cirrhosis)
- Genotype (A, B, C, D)

Centrally measured virus testing results will be used for both the primary endpoint and efficacy endpoints

# 10.3.2. Safety Analyses

Safety analyses will be performed on the SP.

#### Statistical methods

#### Adverse events

All adverse events occurred during the study period will be coded with the latest version of Medical Dictionary for Regulatory Activities (MedDRA) and classified by System Organ Class (SOC) and Preferred Term (PT).

The adverse events, the adverse events causally related with the investigational product, the adverse events resulting in discontinuation of the study, the severe adverse events and the serious adverse events will be summarized, and all the adverse events will be listed.

The frequency and incidence of AE of interest (renal adverse events, hepatic adverse events, and skeletal adverse events) will also be summarized.

# Clinical Laboratory Tests

As for the clinical laboratory values (hematology, clinical chemistry, urinalysis), the summary statistics (number of subjects, mean, median, SD, minimum, maximum) of observed values at each evaluation time point and variation from baseline will be calculated. Shift table from baseline to each evaluation time point will be generated. The measured value for each parameter will be included in the data listings. In addition, subjects found to have test values out of the reference range will be listed.

# Vital Signs

For changes in vital signs (blood pressure, pulse rate, temperature) from baseline to each assessment point, the summary statistics (number of subjects, mean, median, SD, minimum, maximum) will be calculated. The measured value for each parameter will be included in the data listings.
#### **10.3.3.** Interim Analyses

No interim analysis to make statistical investigations will be performed in this study. However, the CRF data by Week 48 will be locked when all subjects (excluding withdrawn subjects) complete Week 48 to collect safety and efficacy data.

#### **10.3.4.** Handling of Withdrawed Subjects

In analyzing the primary endpoint, unless otherwise stated, withdrawed subjects reported during the study period will be treated as non-responders. Other imputation methods will be examined.

#### 11. REFERENCES

Koike K, Suyama K, Ito H, et al. A randomized prospective study showing the non-inferiority of tenofovir to entecavir in treatment-naïve chronic hepatitis B patients. Hepatol Res. 2018;48(1):59-68

Sriprayoon T,Mahidol C,Ungtrakul T, et al. Efficacy and safety of entecavir versus tenofovir treatment in chronic hepatitis B patients: A randomized controlled trial. Hepatol Res. 2017;47(3):E161-E168

Tenozet Tablets 300 mg (Tenofovir Disoproxil Fumarate) Package Insert. Dec 2017.

The Drafting Committee for Hepatitis Management Guidelines, the Japan Society of Hepatology Guidelines for the Management of Hepatitis B Virus Infection (version 3). Aug 2017

Masashi Mizokami, Eiji Tanaka, Kazuaki Chayama, et al. Diagnosis and Treatment of Hepatitis B. Liver. 2010;51:243-60.

# 12. APPENDICES

### **12.1.** Appendix 1: Abbreviations and Trademarks

Abbreviations

| ADV | Adefovir pivoxil |
|-------|--------------------------------------|
| AE | Adverse Event |
| ALP | Alkaline Phosphatase |
| ALT | Alanine Aminotransferase |
| AST | Asparate Aminotransferase |
| CLcr | Creatinine Clearance |
| eCRF | Electronic Case Report Form |
| ETV | Entecavir hydrate |
| eGFR | Estimated Glomerular Filtration Rate |
| FDA | Food and Drug Administration |
| GCP | Good Clinical Practice |
| GSK | GlaxoSmithKline |
| γ-GTP | γ-glutamyltranspeptidase |
| HCC | Hepatocellular carcinoma |
| IEC | Independent Ethics Committee |

# CONFIDENTIAL

# GlaxoSmithKline group of companies

205883

| INR | International Normalized Ratio |
|--------|----------------------------------------------|
| IRB | Institutional Review Board |
| ITT | Intent-To-Treat |
| LAM | Lamivudine |
| MedDRA | Medical Dictionary for Regulatory Activities |
| PCD | Primary completion date |
| PK | Pharmacokinetics |
| PMDA | Pharmaceuticals and Medical Devices Agency |
| PP | Per Protocol |
| PT | Preferred Term |
| RAP | Reporting and Analysis Plan |
| SAE | Serious Adverse Event |
| SD | Standard Deviation |
| SOA | Schedule of Activities |
| SOC | System Organ Class |
| SRM | Study Reference Manual |
| TAF | Tenofovir Alafenamide Fumarate |
| TDF | Tenofovir Disoproxil Fumarate |
| ULN | Upper Limit of Normal |

# Trademark

| Trademarks of the GlaxoSmithKline |
|-----------------------------------|
| group of companies |

| Trademarks not owned by the | |
|------------------------------------|----|
| GlaxoSmithKline group of companies | |
| Tenoze | et |

# 12.2. Appendix 2: Study Governance Considerations

#### **Regulatory and Ethical Considerations**

- This study will be conducted in accordance with the protocol and with:
  - Consensus ethical principles derived from international guidelines including the Declaration of Helsinki and Council for International Organizations of Medical Sciences (CIOMS) International Ethical Guidelines
  - Applicable ICH Good Clinical Practice (GCP) Guidelines
  - The Ordinance on Standards for Conduct of Clinical Trials (MHW Ordinance No. 28 dated March 27, 1997) and applicable laws and regulations regarding quality of medicinal products and medical devices, efficacy and safety assurance, etc.
  - The Ordinance on Good Post-Marketing Study (MHLW Ordinance No.171 dated December 20, 2004)
- The protocol, protocol amendments, ICF, Investigator Brochure, and other relevant documents (e.g., advertisements) must be submitted to an IRB/IEC by the investigator and reviewed and approved by the IRB/IEC before the study is initiated.
- Any amendments to the protocol will require IEC/IRB approval before implementation of changes made to the study design, except for changes necessary to eliminate an immediate hazard to study subjects.
- The investigator will be responsible for the following:
  - Providing written summaries of the status of the study to the IRB/IEC annually or more frequently in accordance with the requirements, policies, and procedures established by the IRB/EC
  - Notifying the IRB/IEC of SAE or other significant safety findings as required by IRB/IEC procedures
  - Providing oversight of the conduct of the study at the site, ICH guidelines, the IRB/IEC, and all other applicable regulations

#### **Financial Disclosure**

Investigators and sub-investigators will provide the sponsor with sufficient, accurate financial information as requested to allow the sponsor to submit complete and accurate financial certification or disclosure statements to the appropriate regulatory authorities. Investigators are responsible for providing information on financial interests during the course of the study and for 1 year after completion of the study.

#### **Informed Consent Process**

Prior to subjects' participation in the study, the investigator (sub-investigator) will fully explain the study using patient information to the subject considered as appropriate or/and to his/her legally authorized representative. During this period, provide the subjects opportunities to ask questions and sufficient time and obtain the consent form signed or signed/sealed dated with the date of consent by the subject and/or his/her legally authorized representative. Subjects may take home the Patient Information/Consent Form to consider about the participation at home. The person who provides explanation and the study collaborator who provides supplemental explanation will sign or sign/seal with the date signed. If a witness is required, the witness should also sign or sign/seal with the date witnessed. The investigator (sub-investigator) will attach the original of the above signed or signed/sealed, and dated Consent Form (and the Patient Information) to the original medical records such as medical chart, retain (follow the storage

regulations of the medical institution, if any), and hand the copy to the subject or his/her legally authorized representative.

- The investigator (sub-investigator) or his/her representative will explain the nature of the study to the subject or his/her legally authorized representative and answer all questions regarding the study.
- Subjects must be informed that their participation is voluntary. The medical record must include a statement that written informed consent was obtained before the subject was enrolled in the study and the date the written consent was obtained. The authorized person obtaining the informed consent must also sign the ICF.
- Subjects must be re-consented to the most current version of the ICF(s) during their participation in the study.
- A copy of the ICF(s) must be provided to the subject or the subject's legally authorized representative.
- Subjects who are rescreened are required to sign a new ICF.

The ICF may contain a separate section that addresses the use of remaining mandatory samples for optional exploratory research in accordance with SOP-GSKF-410. The investigator or authorized designee will explain to each subject the objectives of the exploratory research. Subjects will be told that they are free to refuse to participate and may withdraw their consent at any time and for any reason during the storage period. A separate signature will be required to document a subject's agreement to allow any remaining specimens to be used for exploratory research. Subjects who decline to participate will not provide this separate signature.

#### **Data Protection**

- Subjects will be assigned a unique identifier by the sponsor. Any subject records or datasets that are transferred to the sponsor will contain the identifier only; subject names or any information which would make the subject identifiable will not be transferred.
- The subject must be informed that his/her personal study-related data will be used by the sponsor in accordance with local data protection law. The level of disclosure must also be explained to the subject.
- The subject must be informed that his/her medical records may be examined by Clinical Quality Assurance auditors or other authorized personnel appointed by the sponsor, by appropriate IRB/IEC members, and by inspectors from regulatory authorities.

#### **Publication Policy**

- The results of this study may be published or presented at scientific meetings. If this is
  foreseen, the investigator agrees to submit all manuscripts or abstracts to the sponsor before
  submission. This allows the sponsor to protect proprietary information and to provide
  comments.
- The sponsor will comply with the requirements for publication of study results. In accordance with standard editorial and ethical practice, the sponsor will generally support publication of multicenter studies only in their entirety and not as individual site data. In this case, a coordinating investigator will be designated by mutual agreement.

 Authorship will be determined by mutual agreement and in line with International Committee of Medical Journal Editors authorship requirements.

#### **Dissemination of Clinical Study Data**

Prior to enrolment of subjects, the study information derived from this protocol will be made publicly available on the Clinical Trial Registry System including the website (www.ClinTrials.gov) of the National Institutes of Health (NIH). Where required by applicable regulatory requirements, an investigator signatory will be identified for the approval of the clinical study report. The investigator will be provided reasonable access to statistical tables, figures, and relevant reports and will have the opportunity to review the complete study results at a GSK site or other mutually agreeable location.

GSK will provide the investigator with the full summary of the study results. The investigator will share the summary results with the study subjects, as appropriate.

The results summary will be posted to the GSK Clinical Study Register within 12 months of the PCD or LSLV, whichever is earlier, or any decision to terminate the study. In addition, a manuscript will be submitted to a peer-reviewed journal for publication within 18 months of the LSLV or any decision to terminate the study. When manuscript publication in a peer-reviewed journal is not feasible, further study information will be posted to the GSK Clinical Study Register to supplement the results summary.

#### **Data Quality Assurance**

- All subject data relating to the study will be recorded on electronic CRF (eCRF) unless
  transmitted to the sponsor or designee electronically (e.g., laboratory data). The investigator
  is responsible for verifying that data entries are accurate and correct by physically or
  electronically signing the CRF.
- The investigator must maintain accurate documentation (source data) that supports the information entered in the CRF.
- The investigator must permit study-related monitoring, audits, IRB/IEC review, and regulatory agency inspections and provide direct access to source data documents.
- The sponsor or designee is responsible for the data management of this study including quality checking of the data.
- Study monitors will perform ongoing source data verification to confirm that data entered
  into the CRF by authorized site personnel are accurate, complete, and verifiable from source
  documents; that the safety and rights of subjects are being protected; and that the study is
  being conducted in accordance with the latest approved protocol and any other study
  agreements, ICH, GCP, and all applicable regulatory requirements.
- Records and documents, including signed ICF, pertaining to the conduct of this study must
  be retained by the investigator for 25 years from the issue of the final Clinical Study Report
  (CSR)/ equivalent summary unless local regulations or institutional policies require a longer
  retention period. No records may be destroyed during the retention period without the written
  approval of the sponsor. No records may be transferred to another location or party without
  written notification to the sponsor.

#### **Source Documents**

- Source documents provide evidence for the existence of the subject and substantiate the integrity of the data collected. Source documents are filed at the investigator's site.
- Data reported on the CRF or entered in the eCRF that are transcribed from source documents
  must be consistent with the source documents or the discrepancies must be explained. The
  investigator may need to request previous medical records or transfer records, depending on
  the study. In addition, current medical records must be available.
- Definition of what constitutes source data can be found in the source document correspondence list.

#### Study and Site Closure

GSK or its designee reserves the right to close the study site or terminate the study at any time for any reason at the sole discretion of GSK. Study sites will be closed upon study completion. A study site is considered closed when all required documents and study supplies have been collected and a study-site closure visit has been performed.

The investigator may initiate study-site closure at any time, provided there is reasonable cause and sufficient notice is given in advance of the intended termination.

Reasons for the early closure of a study site by the sponsor or investigator may include but are not limited to:

- Failure of the investigator to comply with the protocol, the requirements of the IRB/IEC or local health authorities, the sponsor's procedures, or GCP guidelines
- Inadequate recruitment of subjects by the investigator
- Discontinuation of marketing of the investigational product

#### **Study Period**

August 2017 to December 2019

#### Implementation system

Attachment 1 provides the sponsor information. Attachment 2 provides a list of medical institutions and investigators.

# **12.3.** Appendix 3: Adverse Events: Definitions and Procedures for Recording, Evaluating, Follow-up, and Reporting

#### **Definition of AE**

#### AE Definition

- An AE is any untoward medical occurrence in a clinical study subject, temporally
  associated with the use of a study treatment, whether or not considered related to the study
  treatment.
- NOTE: An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study treatment.

#### **Events Meeting the AE Definition**

- Any abnormal laboratory test results (hematology, clinical chemistry, or urinalysis) or other safety assessments (e.g., ECG, radiological scans, vital signs measurements), including those that worsen from baseline, considered clinically significant in the medical and scientific judgment of the investigator (i.e., not related to progression of underlying disease).
- Exacerbation of a chronic or intermittent pre-existing condition including either an increase in frequency and/or intensity of the condition.
- New conditions detected or diagnosed after study treatment administration even though it
  may have been present before the start of the study.
- Signs, symptoms, or the clinical sequelae of a suspected drug-drug interaction.
- Signs, symptoms, or the clinical sequelae of a suspected overdose of either study treatment
  or a concomitant medication. Overdose per se will not be reported as an AE/SAE unless it is
  an intentional overdose taken with possible suicidal/self-harming intent. Such overdoses
  should be reported regardless of sequelae.
- "Lack of efficacy" or "failure of expected pharmacological action" per se will not be reported as an AE or SAE. Such instances will be captured in the efficacy assessments. However, the signs, symptoms, and/or clinical sequelae resulting from lack of efficacy will be reported as AE or SAE if they fulfil the definition of an AE or SAE.

#### Events **NOT** Meeting the AE Definition

- Any clinically significant abnormal laboratory findings or changes in other safety
  assessments which are associated with the underlying disease, unless judged by the
  investigator to be more severe than expected for the subject's condition.
- The disease/disorder being studied or expected progression, signs, or symptoms of the disease/disorder being studied, unless more severe than expected for the subject's condition.
- Medical or surgical procedure (e.g., endoscopy, appendectomy): the condition that leads to the procedure is the AE.
- Situations in which an untoward medical occurrence did not occur (social and/or convenience admission to a hospital).
- Anticipated day-to-day fluctuations of pre-existing disease(s) or condition(s) present or detected at the start of the study that do not worsen.

#### 205883

#### **Definition of SAE**

If an event is not an AE per definition above, then it cannot be an SAE even if serious conditions are met (e.g., hospitalization for signs/symptoms of the disease under study, death due to progression of disease).

#### A SAE is defined as any untoward medical occurrence that, at any dose:

#### a. Results in death

#### b. Is life-threatening

The term 'life-threatening' in the definition of 'serious' refers to an event in which the subject was at risk of death at the time of the event. It does not refer to an event, which hypothetically might have caused death, if it were more severe.

# c. Requires inpatient hospitalization or prolongation of existing hospitalization

In general, hospitalization signifies that the subject has been detained (usually involving at least an overnight stay) at the hospital or emergency ward for observation and/or treatment that would not have been appropriate in the physician's office or outpatient setting. Complications that occur during hospitalization are AEs. If a complication prolongs hospitalization or fulfills any other serious criteria, the event is serious. When in doubt as to whether "hospitalization" occurred or was necessary, the AE should be considered serious.

Hospitalization for elective treatment of a pre-existing condition that did not worsen from baseline is not considered an AE.

## d. Results in persistent disability/incapacity

- The term means a substantial disruption of a person's ability to conduct normal life functions.
- This definition is not intended to include experiences of relatively minor medical significance such as uncomplicated headache, nausea, vomiting, diarrhea, influenza, and accidental trauma (e.g., sprained ankle) which may interfere with or prevent everyday life functions but do not constitute a substantial disruption.

#### e. Is a congenital anomaly/birth defect

#### f. Other situations:

• Medical or scientific judgment should be exercised in deciding whether SAE reporting is appropriate in other situations such as important medical events that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the subject or may require medical or surgical intervention to prevent one of the other outcomes listed in the above definition. These events should usually be considered serious. Examples of such events include invasive or malignant cancers, intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias or convulsions that do not result in hospitalization, or development of drug dependency or drug abuse.

#### g. Events meeting liver chemistry stopping criteria

- Bilirubin  $\geq 2$  times ULN and >35% direct bilirubin
- International Normalized Ratio (INR) > 1.5 in absence of warfarin
- Evidence of clinical decompensation (development of encephalopathy, ascites, hypoalbuminea [albumin ≤ 3g/dL]), or variceal bleeding
- ALT ≥ 20 times ULN in the absence of increased bilirubin or evidence of clinical decompensation, if persisting ≥ 2 weeks or accompanied by worsening hepatitis symptoms

#### **Definition of Cardiovascular Events**

#### Cardiovascular Events (CV) Definition:

Investigators will be required to fill out the specific CV event page of the CRF for the following AEs and SAEs:

- Myocardial infarction/unstable angina
- Congestive heart failure
- Arrhythmias
- Valvulopathy
- Pulmonary hypertension
- Cerebrovascular events/stroke and transient ischemic attack
- Peripheral arterial thromboembolism
- Deep venous thrombosis/pulmonary embolism
- Revascularization

### **Recording AE and SAE**

#### AE and SAE Recording

- When an AE/SAE occurs, it is the responsibility of the investigator to review all
  documentation (e.g., hospital progress notes, laboratory, and diagnostics reports) related to
  the event.
- The investigator will then record all relevant AE/SAE information in the CRF.
- It is **not** acceptable for the investigator to send photocopies of the subject's medical records to GSK in lieu of completion of the GSK /AE/SAE CRF page.
- There may be instances when copies of medical records for certain cases are requested by GSK. In this case, all subject identifiers, with the exception of the subject number, will be redacted on the copies of the medical records before submission to GSK.
- The investigator will attempt to establish a diagnosis of the event based on signs, symptoms, and/or other clinical information. Whenever possible, the diagnosis (not the individual signs/symptoms) will be documented as the AE/SAE.

#### **Assessment of Intensity**

The investigator will make an assessment of intensity for each AE and SAE reported during the study and assign it to one of the following categories:

- Mild: An event that is easily tolerated by the subject, causing minimal discomfort and not interfering with everyday activities.
- Moderate: An event that causes sufficiently discomfort and interferes with normal everyday activities.
- Severe: An event that prevents normal everyday activities. An AE that is assessed as severe
  should not be confused with an SAE. Severity is a category utilized for rating the intensity
  of an event; and both AE and SAE can be assessed as severe.

An event is defined as 'serious' when it meets at least 1 of the predefined outcomes as described in the definition of an SAE, NOT when it is rated as severe.

#### Assessment of Causality

• The investigator is obligated to assess the relationship between study treatment and each occurrence of each AE/SAE.

- A "reasonable possibility" of a relationship conveys that there are facts, evidence, and/or arguments to suggest a causal relationship, rather than a relationship cannot be ruled out.
- The investigator will use clinical judgment to determine the relationship.
- Alternative causes, such as underlying disease(s), concomitant therapy, and other risk
  factors, as well as the temporal relationship of the event to study treatment administration
  will be considered and investigated.
- The investigator (sub-investigator) will also consult the Investigator's Brochure (IB) and/or Product Information, for marketed products, in his/her assessment.
- For each AE/SAE, the investigator <u>must</u> document in the medical notes that he/she has reviewed the AE/SAE and has provided an assessment of causality.
- There may be situations in which an SAE has occurred and the investigator has minimal
  information to include in the initial report to GSK. However, it is very important that the
  investigator always make an assessment of causality for every event before the initial
  transmission of the SAE data to GSK.
- The investigator may change his/her opinion of causality in light of follow-up information and send an SAE follow-up report with the updated causality assessment.
- The causality assessment is one of the criteria used when determining regulatory reporting requirements.

#### Follow-up of AE and SAE

- The investigator is obligated to perform or arrange for the conduct of supplemental
  measurements and/or evaluations as medically indicated or as requested by GSK to
  elucidate the nature and/or causality of the AE or SAE as fully as possible. This may include
  additional laboratory tests or investigations, histopathological examinations, or consultation
  with other health care professionals.
- If a subject dies during participation in the study or during a recognized follow-up period, the investigator will provide GSK with a copy of any post-mortem findings including histopathology.
- New or updated information will be recorded in the originally completed CRF.
- The investigator will submit any updated SAE data to GSK within 24 hours of receipt of the information.
- Any updated data on non-SAEs considered associated with the use of study treatment in the
  post-marketing study will be submitted by the investigator to GSK within 24 hours of
  receipt of the information.

#### Reporting of SAE to GSK

#### SAE Reporting to GSK via eCRF

- The primary mechanism for reporting SAE to GSK will be the eCRF.
- If the electronic system is unavailable for more than 24 hours, then the site will use the paper SAE data collection tool (see next section).
- The site will enter the SAE data into the electronic system as soon as it becomes available.
- The investigator or medically-qualified sub-investigator must show evidence within the eCRF (e.g., check review box, signature, etc.) of review and verification of the relationship of each SAE to IP/study participation (causality) within 72 hours of SAE entry into the eCRF.

- After the study is completed at a given site, the eCRF will be taken off-line to prevent the entry of new data or changes to existing data.
- If a site receives a report of a new SAE from a study subject or receives updated data on a previously reported SAE after the eCRF has been taken off-line, then the site can report this new or updated information on a paper SAE form (see next section) or to the sponsor's medical monitor/study contact by telephone.
- Contacts for SAE reporting can be found in Attachment 1.
- The non-SAEs considered associated with the use of study treatment in the post-marketing clinical study should be reported in the same manner.

# SAE Reporting to GSK via Paper CRF

- Facsimile transmission of the SAE paper CRF is the preferred method to transmit this information to the sponsor's **medical monitor or the SAE coordinator**.
- In rare circumstances and in the absence of facsimile equipment, notification by telephone is acceptable with a copy of the SAE pages of the CRF sent by overnight mail or courier service
- Initial notification via telephone does not replace the need for the investigator to complete and sign the SAE CRF pages within the designated reporting time frames.
- Contacts for SAE reporting can be found in Attachment 1.
- The non-SAEs considered associated with the use of study treatment in the post-marketing clinical study should be reported in the same manner.

### 12.4. Appendix 4: Contraceptive Guidance and Collection of Pregnancy Information

#### **Definitions**

### Woman of Childbearing Potential (WOCBP)

A woman is considered fertile following menarche and until becoming post-menopausal unless permanently sterile (see below)

#### Women in the following categories are not considered WOCBP

- 1. Premenarchal
- 2. Premenopausal female with ONE of the following:
  - Documented hysterectomy
  - Documented bilateral salpingectomy
  - Documented bilateral oophorectomy

Note: Documentation can come from the site personnel's review of subject's medical records, medical examination, or medical history interview.

#### 3. Postmenopausal female

- A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy (HRT). However, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient.
- Females on HRT and whose menopausal status is in doubt will be required to use one of
  the non-hormonal highly effective contraception methods if they wish to continue their
  HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of
  postmenopausal status before study enrolment.

#### **Contraception Guidance**

#### Female subjects

Female subjects of childbearing potential are eligible to participate if they agree to use a highly effective method of contraception consistently and correctly as described in Table 4.

#### Table 4 Highly effective contraception methods

#### Highly Effective Contraceptive Methods That Are User Dependent a

Failure rate of <1% per year when used consistently and correctly.

Combined (estrogen- and progestogen-containing) hormonal contraception associated with inhibition of ovulation<sup>b</sup>

• Oral

#### Highly Effective Methods That Are User Independent

- Intrauterine device (IUD)
- Intrauterine hormone-releasing system (IUS)

### Vasectomized partner

(A vasectomized partner is a highly effective contraception method provided that the partner is the sole male sexual partner of the WOCBP and the absence of sperm has been confirmed. If not, an additional highly effective method of contraception should be used.)

#### Sexual abstinence

(Sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study drug. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the study and the preferred and usual lifestyle of the subject.)

#### NOTES:

- a. Typical use failure rates may differ from those when used consistently and correctly. Use should be consistent with local regulations regarding the use of contraceptive methods for subjects in clinical studies.
- b. Hormonal contraception may be susceptible to interaction with the study treatment, which may reduce the efficacy of the contraceptive method. In this case, two highly effective methods of contraception should be utilized during the treatment period and for at least 4 days after the last dose of study treatment.

#### **Pregnancy Testing**

- WOCBP should only be included after a confirmed menstrual period and a negative highly sensitive urine pregnancy test.
- Additional pregnancy testing is not required during the treatment and after the last dose of study treatment and as required locally.
- Pregnancy testing will be performed whenever a menstrual cycle is missed or when pregnancy is otherwise suspected.
- Pregnancy testing will be performed using the test kit approved by the sponsor and in accordance with instructions provided in its package insert.

# Collection of Pregnancy Information

# Female Subjects who become pregnant

- Investigator will collect pregnancy information on any female subject, who becomes pregnant while participating in this study.
- Information will be recorded on the appropriate form and submitted to GSK within 24 hours of learning of a subject's pregnancy.
- Subject will be followed to determine the outcome of the pregnancy. The investigator will collect follow up information on subject and neonate, which will be forwarded to GSK Generally, follow-up will not be required for longer than 6 to 8 weeks beyond the estimated delivery date.
- Any termination of pregnancy will be reported, regardless of fetal status (presence or absence of anomalies) or indication for procedure.
- While pregnancy itself is not considered to be an AE or SAE, any pregnancy complication or elective termination of a pregnancy will be reported as an AE or SAE.
- A spontaneous abortion is always considered to be an SAE and will be reported as such.
- Any SAE occurring as a result of a post-study pregnancy which is considered reasonably related to the study treatment by the investigator, will be reported to GSK as described in Appendix 3. While the investigator is not obligated to actively seek this information in former study subjects, he or she may learn of an SAE through spontaneous reporting.

Any female subject who becomes pregnant while participating

• Will be withdrawn from the study

# **12.5.** Appendix 5: Liver Safety: Required Actions and Follow-up Assessment and Study Treatment Rechallenge Guidelines

Liver chemistry stopping and follow-up assessment criteria in phase III-IV studies will be specified in order to secure the safety of the subjects and evaluate the etiology of liver events.

# Liver chemistry stopping criteria and required follow-up assessment in phase III-IV studies

| | Liver chemistry stopping criteria | | | |
|---|---|---|---|---|
| <b>Bilirubin¹</b> Bilirubin ≥ 2 times ULN and >35 | | | | direct bilirubin |
| | INR <sup>1</sup> | INR > 1.5 in absence of warfarin | | |
| Sy | mptoms | Evidence of clinical decompensation (development of encephalopathy, ascites, | | |
| | hypoalbuminea [albumin ≤ 3g/dI | | | or variceal bleeding |
| | | ALT ≥ 20 times ULN in the abse | ence | of increased bilirubin or evidence of clinical |
| | | decompensation, if persisting $\geq 2$ | 2 we | eks or accompanied by worsening hepatitis |
| | | symptoms | | |
| | | Required actions and | live | r event endpoints |
| | A | ctions to be taken | | Liver event endpoints |
| • | Discontinu | ie study treatment immediately | • | Serum testing <sup>2</sup> related to virus hepatitis |
| • | Report the | information to the sponsor | • | Measure the INR and monitor each liver |
| | within 24 | hours. | | function test value until decreasing trend is |
| | | t meets SAE criteria as well, | | observed in transaminase levels. |
| | | 3 | • | Only the subjects who were complicated |
| | Event" and "SAE" sections of the CRF. <sup>1</sup> | | | with CHB at the time of enrolment |
| | • Investigate the liver event endpoints (refer | | | (confirmed by positive hepatitis B surface |
| | to the right column for endpoints). | | | antigen (HBsAg)): HBV-DNA quantitative |
| | • Subjects will be followed up until the liver | | | analysis |
| | function test value becomes normal, | | • | Obtain blood sample for PK analysis |
| | stabilizes or returns to the baseline level | | | within 24 hours after the last dose. <sup>3</sup> |
| (refer to the "Follow-up assessment" | | • | Serum creatine phosphokinase (CPK) and | |
| below). | | | lactate dehydrogenase (LDH) | |
| | _ | treatment must not be re- | • | Fractionate bilirubin, if total bilirubin $\ge 2 \text{ x}$ |
| | initiated/r | re-administered to subjects. | | ULN |
| | | | • | Obtain blood count including WBC |
| Falla | w-up asse | ssment. | _ | differential to assess eosinophilia |
| | - | | • | Record the occurrence and worsening of clinical symptoms <sup>4</sup> of hepatic impairment |
| <ul><li>Bilirubin or INR Criteria:</li><li>The liver function tests (ALT, AST, ALP,</li></ul> | | | or hypersensitivity on the AE CRF. | |
| bilirubin) should be performed again | | • | Record use of concomitant medications | |
| within 24 hours and liver event endpoints | | | including acetaminophen, herbal remedies, | |
| will be examined (refer to the right column | | | and other over the counter medications on | |
| | for endpoi | nts). | the concomitant medications CRF. | |
| • | Follow-up | will be performed twice a week | • | Record alcohol intake on the liver event |
| | until the li | ver function test value becomes | | CRF. |
| | normal, sta | abilizes or returns to the baseline | | |
| | level. | | | |

 Complete the liver imaging and/or liver biopsy CRFs if these tests are performed.

#### Other criteria:

- Subjects with ALT ≥ 20 times ULN who otherwise do not meet other stopping criteria outlined above can continue study medication, but should be monitored weekly.
- If, after 2 weeks of monitoring, ALT < 20 times ULN, subjects should be monitored twice monthly until the liver function test value becomes normal, stabilizes or returns to the baseline level. However, if during the monitoring period, subjects meet the liver chemistry threshold stopping criteria or are unable to return for weekly follow-up, investigational product must be stopped and follow-up will be performed until the liver function test value becomes normal, stabilizes or returns to the baseline level.

- HBV-DNA level resistance analysis (only in the subject who has shown virological breakthrough)
- HBeAg/Ab
- Prothrombin time

#### Bilirubin or INR criteria:

- Quantitative determinations of antinuclear antibody, antismooth muscle antibody, anti-liver/kidney microsome antibody type I and immunoglobulin G (IgG) or gammaglobulin
- Perform liver imaging (ultrasound, magnetic resource, or computerized tomography) and/or liver biopsy to evaluate liver disease and record on the liver event CRF.
- Events indicating severe liver injury (possible Hy's Law) (bilirubin ≥ 2 times ULN and >35% direct bilirubin, or INR > 1.5 in the absence of warfarin) must be reported as an SAE.
- 2. Hepatitis A IgM antibody, hepatitis B surface antigen (HBsAg) and hepatitis B core antibody (IgM), hepatitis C RNA, cytomegalovirus IgM antibody, Epstein-Barr virus capsid antigen IgM antibody (if not feasible, perform the heterophile agglutination test), hepatitis E IgM antibody or hepatitis E RNA
- 3. Record the date/time of the PK blood sample draw and the date/time of the last dose of investigational product prior to blood sample draw on the CRF. If the date or time of the last dose is unclear, provide the subject's best approximation. If the date/time of the last dose cannot be approximated OR a PK sample cannot be collected in the time period indicated above, do not obtain a PK sample. Refer to the Study Reference Manual (SRM) for procedures for handling and transferring samples.
- 4. Symptoms considered to be related to liver impairment (fatigue, nausea, vomiting, right upper quadrant pain or tenderness, jaundice, etc.), or symptoms considered to be related to hypersensitivity (fever, rash, eosinophilia, etc.).

#### References

James LP, Letzig L, Simpson PM, Capparelli E, Roberts DW, Hinson JA, Davern TJ, Lee WM. Pharmacokinetics of Acetaminophen-Adduct in Adults with Acetaminophen Overdose and Acute Liver Failure. Drug Metab Dispos 2009; 37:1779-1784.

Le Gal F, Gordien E, Affolabi D, Hanslik T, Alloui C, Dény P, Gault E. Quantification of Hepatitis Delta Virus RNA in Serum by Consensus Real-Time PCR Indicates Different Patterns of

# 2017N312381\_06 CONFIDENTIAL

# GlaxoSmithKline group of companies

205883

Virological Response to Interferon Therapy in Chronically Infected Patients. J Clin Microbiol. 2005;43(5):2363–2369.

#### 205883

## 12.6. Appendix 6: Prohibited Drugs

Prohibit the use of the below drugs from the initiation of the study treatment:

- Interleukin-2 preparations
- Ursodeoxycholic acid preparations
- Herbal medicine with positive effects on hepatic dysfunction
- Antiviral drugs with an inhibitory effect on HBV growth (excluding ADV and TAF, which should be prohibited from the day of the informed consent)

TDF is prohibited from the day of the consent until the day before the initiation of the study treatment (TDF will be administered as an investigational product from Day 1)

Prohibit the use of the below drugs from the day of the informed consent:

- Other investigational products
- Interferon preparations
- HB vaccine therapy
- Glucocorticoid preparations (excluding topical preparations such as ointment and cream)
- Immunosuppressants (e.g., azathioprine and cyclophosphamide) or chemotherapeutic agents (e.g., etoposide) (excluding topical preparations such as ointment and cream)
- Drugs influential on the renal functions shown below (excluding topical preparations such as ointment and cream)
  - Nephrotoxic drugs (e.g., aminoglycoside-class antibiotics, amphotericin B, vancomycin, foscarnet, cisplatin, pentamidine, tacrolimus, cyclosporine, some contrast media [ionic high osmolar contrast medium, ionic low osmolar contrast media])
  - Drugs competing in renal excretion (excluding temporary use, e.g., probenecid)

Prohibit the use of the below drugs influential on the renal functions within 7 days prior to initiation of the study treatment:

• Overdose NSAIDs (excluding temporary or topical use)

# 12.7. Appendix 7: Evaluation of Baseline Values

#### 12.7.1. Participant Backgrounds

At the time of screening, the following items will be examined and recorded in the eCRF.

- Birth year, gender, race
- Time of diagnosis of CHB/cirrhosis B
- Cardiovascular history/risk factors
- History related to liver disease
- Complications
- Name of the drug for the treatment of CHB and treatment period within 2 years
- History of alcohol consumption and smoking
- Family history of cardiovascular risk factors
- Measured values at 2 time points (with an interval of at least 3 months, and at least one point
  within 1 year from screening) for subjects in whom changes in HBsAg before screening can
  be confirmed.

# 12.7.2. Diagnosis of Cirrhosis B

Cirrhosis will be diagnosed when applicable to either of the following.

- A case where definite diagnosis of cirrhosis has been made by liver biopsy or abdominoscopy performed within one year before obtaining consent
- A case where cirrhosis can be diagnosed in clinical overall diagnosis including abdominal imaging tests (ultrasonography, CT, MRI, etc.) (see Table 5)

| | Test item | Criterion |
|---|---|---|
| Hematology | Platelet count | $\leq 120,000 / \mu L$ |
| Clinical Chemistry | Hyaluronate level | ≥ 100 ng/mL |
| Abdominal imaging test <sup>2</sup> | Ultrasonography, CT, MRI, etc. | <ol> <li>Concavity and convexity<br/>on the liver surface</li> <li>Echo pattern changes in<br/>the hepatic parenchyma</li> <li>Findings of portal<br/>hypertension</li> </ol> |

Table 5 Cirrhosis diagnosis criteria<sup>1</sup>

- 1. Cirrhosis is diagnosed when all the criteria are met. Use the results of hematology, clinical chemistry and abdominal imaging test obtained at the time of screening.
- 2. One of the criteria 1 to 3 must be met for abdominal imaging tests.

#### 12.7.3. Bone densitometry

Perform densitometry on either lumbar spine or femur, using DEXA (refer to Table 6). If there is a difficulty to perform with DEXA or on either lumbar spine or femur, other region (radius or calcaneus) or other method (SEXA or ultrasound) may be selected.

Table 6 Region to perform bone densitometry

| | Preferred | Substitute | |
|--------|-----------|------------|------------|
| Method | DEXA | SEXA | Ultrasound |

205883

| Region | lumbar spine radius | | calcaneus |
|--------|------------------------|-----------|-----------|
| | femur | calcaneus | |
| | radius <sup>1</sup> | | |
| | calcaneus <sup>1</sup> | | |

<sup>1.</sup> Measure this region if the lumbar spine or femur is not available

If densitometry is required during the study or at study completion/discontinuation, use the same method and region performed at baseline.